# Target ADHD Executive Working Memory Training Replication Study

Study Protocol

IRB Approval Date: 9/22/2023

## Behavioral and Neural Target Engagement for ADHD Executive Working Memory Training

### Phase II

This proposal is based on converging evidence that suggests prior ADHD working memory training studies might have produced lackluster clinical outcomes because they focused on enhancing the wrong cognitive and neurobiological targets. The proposed study will replicate target engagement as assessed in the first phase while also determining if it correlates with clinically meaningful improvements in ADHD dysfunction. The full project was designed so that if these study aims are successful, the data we obtain will be adequate to support a future preliminary efficacy clinical trial.

Many investigators have attempted to show that using intensive cognitive training to increase Attention-Deficit/Hyperactivity Disorder (ADHD) patients' capacity to store information within WM might also reduce symptom severity or functional impairment. Those studies were based on strong evidence for WM behavioral and neural dysfunction in ADHD, a widely-held belief that WM-related brain dysfunction is etiologically significant, and arguments that impaired WM contributes to the maintenance of the disorder. But despite promising early evidence for WM storage training potential efficacy, a decade of equivocal and negative outcomes from several well-designed randomized clinical trials have left investigators wondering why meaningful, replicable ADHD clinical improvements are not always achieved when WM storage capacity is reliably enhanced. Because few investigators want to mistakenly abandon such a promising intervention premise, there is a search for novel working memory-related treatment targets that focus on something other than simple WM storage capacity. In this proposal, we synthesize published findings and provide our own pilot neuroimaging evidence to argue that a better WM training target might be brain regions that specifically underlie the executive aspects of WM. Such executive working (EWM) memory operations represent patients' ability to effectively use the information represented in WM for behavioral and cognitive control. These abilities likely are more meaningful to ADHD behavioral impairment than merely how large patients' general WM storage capacity is. An extensive theoretical framework supports that the 'working' part of WM involves a small handful of discrete cognitive operations that flexibly manipulate information within WM, or stabilize WM representations in the face of different types of environmental distraction. Dozens of prior fMRI studies reliably link the four primary types of these EWM operations to activity within specific brain regions – the superior frontal sulcus and mid-lateral prefrontal cortex. Converging evidence including our pilot evidence shows these regions function abnormally in ADHD, predict ADHD symptom severity, and can be enhanced by practicing EWM tasks. NIMH's R61/R33 experimental therapeutics mechanism is ideal to learn if a typical 5week, course of intensive training that uses these EWM exercises can engage the proposed brain targets linked to both EWM ability and to ADHD dysfunction. As the neuroscience-guided, initial 2-year R61 study phase achieved its milestones, this R33 study phase will seek to replicate, and then show the relevance of target engagement to ADHD clinical function. If both R61/R33 aims are achieved, a series of secondary analyses will re-examine the trial outcome data. These efforts will inform the design of any subsequent preliminary efficacy study, facilitating a rapid transition into larger-scale efficacy testing.

Over a decade ago, considerable interest emerged in whether intensive practice of working memory (WM) tasks designed to expand one's overall capacity to store information briefly in mind might benefit patients with Attention-Deficit/Hyperactivity Disorder (ADHD). WM training has a convincing neuroscientific foundation and there was exciting preliminary evidence that prompted WM training intervention development. Nearly all clinical trials to date that have focused on increasing simple short-term WM storage capacity have been disappointing. Investigators remain perplexed why ADHD patients make very reliable, usually persistent WM gains, but simply having a larger WM capacity does not convincingly result in ADHD symptom improvements. Our pilot studies suggest WM training might live up to early expectations if investigators switch focus to a new training target – 'executive working memory' (EWM). EWM refers to a few selective attention-based cognitive processes that operate within WM either to flexibly allow information to be manipulated, or to stabilize and protect mental representations when they are needed to guide behavior. Converging evidence supports EWM as a potentially better training target than WM storage capacity. Importantly, our pilot data also show EWM practice alters ADHD brain function in regions linked to ADHD symptom severity in our prior research. This proposal includes a 2-year milestone-driven R61 initial test of target engagement using a new EWM training intervention in n=62ADHD-diagnosed adolescents randomized to a 'sham training' placebo or to train on 4 different EWM tasks per session 4 times each week. Exercise difficulty levels in the active intervention increased across 5 weeks to continually challenge EWM ability. EWM training used a novel, remotely-supervised 'at home' computerized training approach. Since the R 61 EWM training target engagement milestones were met, a 3-year R33 phase will begin. The R33 will replicate target engagement in another randomized placebo-controlled trial of *n*=90 new ADHD adolescents and attempt to establish a convincing link between the hypothesized targets and ADHD symptom expression. It also will characterize ADHD brain activity or EWM ability changes relative to typical levels seen in an *n*=40 non-ADHD control group.

**R33 AIM 1 Replicate and Extend ADHD EWM Training Target Engagement Relative to Placebo** Another randomized, placebo-controlled trial of *n*=90 new ADHD adolescents will provide evidence needed to support a subsequent efficacy trial – replication of target engagement and confirmation of clinical relevance.

R33 Hypotheses 1-2 Compared to a 'sham training' placebo for which we expect no EWM target change:

- 1) We will replicate both SFS/mid-latPFC brain activity/connectivity and behavioral changes seen in the R61.
- 2) We will see evidence of 'near transfer' of EWM behavioral training gains to non-trained EWM tests.

R33 AIM 2 Establish a Link Between Target Engagement and ADHD Symptom Expression

Data will be used to test assumptions the proposed neural targets are relevant to ADHD clinical impairment.

R33 Hypotheses 3-4 There will be a significant association between EWM engagement and ADHD symptoms:

- 3) Before training, ADHD symptom severity will correlate with EWM brain function and behavior (r > .35).
- 4) The degree of fMRI-measured EWM training target engagement will significantly correlate with ADHD outcome measured by ADHD symptom severity rating scales and secondary functional inventories.

Unmet ADHD Treatment Need DSM 5 Attention-Deficit/Hyperactivity Disorder (ADHD) <sup>1</sup> affects 5-7% of children and adolescents <sup>2-4</sup>. It is marked by excessive impulsivity/hyperactivity and inattention causing significant academic <sup>5-11</sup>, employment, legal or psychosocial problems and risk for other psychopathology and substance disorder <sup>7, 12, 13</sup> despite the best-supported treatments <sup>14-16</sup>. Stimulant-based medications are first-line recommended ADHD treatments <sup>17</sup>, but have meaningful limitations. Medications manage immediate problem behavior, but do not prevent poorer ADHD long-term educational, vocational, or social outcomes <sup>18-24</sup>. Roughly <sup>1</sup>/<sub>4</sub> of ADHD patients fail to show any beneficial response <sup>25</sup>. Medications can be very unpopular with some patients and their parents <sup>26, 27</sup> due to intolerance of side effects <sup>28, 29</sup> or parental concerns of misuse <sup>30-33</sup> from a high abuse potential <sup>30-32, 34</sup> and fears about growth and health risks <sup>35, 36</sup>. Only about half of ADHD-diagnosed children <sup>37</sup> and adolescents <sup>38</sup> use medications. As such, at least half of ADHD patients could benefit from an effective alternative, non-pharmacological treatment to help reduce the \$143-266 billion annual estimated economic burden of ADHD in the U.S. from healthcare costs, lost workforce productivity, and similar factors <sup>39</sup>. An effective alternative ideally would not be another temporary palliative, but instead offer sustained benefits.

Why Train Working Memory to Treat ADHD? Over the past decade, considerable effort has been poured into studying a non-pharmacological cognitive training approach for ADHD that seeks to improve working memory (WM) through weeks of continually challenging training sessions. Such approaches are based upon a well-supported premise that intensive practice reliably induces long-term synaptic connectivity and brain structure changes 40-42 (i.e., experience-dependent 'neuroplasticity') in networks that underlie the specific ability that has been trained <sup>43-51</sup>. A strong appeal of cognitive training is that it might offer enduring therapeutic benefits for ADHD patients from neuroplastic changes - particularly if those changes occur early to optimize neurodevelopmental trajectories into adulthood. The ultimate goal of these intervention development efforts has always been to reduce ADHD symptom severity and associated clinical dysfunction. The premise of WM training for ADHD rests on a reasonable conceptual foundation that links WM performance on brief WM information storage tasks to attention abilities 40, 52, 53, general aptitude (IQ 54-56, reasoning ability 57, or SAT performance 58), and academic achievement 54, 58-64. Moreover, ADHD patients' performance on some WM tasks predicts 'real world' ADHD-like behaviors in non-ADHD persons 65, 66, e.g., multi-tasking 67, 68, mind wandering 69, and following directions 70, 71. Meta-analyses of neuropsychological studies also show WM deficits are among the most consistently found cognitive impairments in ADHD 72-75. It has been proposed that WM training might work by directly remediating WM-related ADHD brain dysfunction believed to be etiologically-significant for the disorder <sup>72, 76-84</sup>. Not only is WM a proposed endophenotype for common genetic risk in ADHD <sup>85, 86</sup>, recent studies have begun to demonstrate WM's etiological importance by showing ADHD patients' WM ability levels mediate links between ADHD polygenic risk scores and ADHD symptom expression 85,87 in ways not found for other cognitive deficits 88. In the WM training earliest studies, pioneering approaches (e.g., Cogmed™) were found not only to increase ADHD WM storage capacity on behavioral tests, but in non-ADHD also to alter grey and white matter brain structure, dopaminergic function, and brain activity 89. Indeed, numerous fMRI studies of young 90-94 and older adults 90, 95, and fMRI 91, 96, 97 and EEG 98 functional connectivity studies done after WM training show brain network 99-102 connectivity reconfiguration and strengthening within the frontoparietal system engaged for WM, and with key WM-specialized regions in other parts of the brain. As such, there was great excitement we ultimately might find these neural effects converged with evidence for WM-related brain dysfunction that has been found in ADHD in over a dozen fMRI studies 103-106.

**WM Storage Training Fails Expectations** Nearly all ADHD WM training research to date has focused on increasing WM storage capacity. These efforts have fallen short of expectations. On the one hand, qualitative <sup>107-113</sup> and meta-analytic <sup>114-117</sup> reviews conclude WM training reliably improves ADHD WM capacity, with gains that persist over time <sup>118-120</sup>. Disappointingly however, the evidence these WM capacity gains translate into improved ADHD symptom severity or better functioning is marginal and inconsistent. The earliest clinical trials found improved parent-, teacher-, or self-rated ADHD severity <sup>53, 121-125</sup> or objectively-measured ADHD behavior (e.g., actigraph-measured motor restlessness or classroom time-on-task <sup>53, 126</sup>), with some evidence that gains might persist for months <sup>53, 123, 125</sup>. However, this evidence came almost entirely from 'open label' trials where expectancy effects typically inflate perception of clinical benefit. Subsequent, better-designed randomized clinical trials (RCTs) have not strongly supported WM storage training efficacy in ADHD. While several RCTs found WM training can produce modest clinical improvement, WM training groups typically do not outperform active treatment control groups. A recent meta-analysis has concluded RCT blinding reduces the promising effects seen in the earlier open label trials to clinically insignificant levels <sup>127</sup>. Perplexingly, those RCTs often failed to replicate the same small positive outcomes <sup>107, 125, 126, 128</sup>. By and large, efforts to train other executive

abilities (e.g., response inhibition, sustained attention, etc.) (e.g., <sup>129, 130</sup>; see meta-analysis <sup>116</sup>), or to train several executive abilities together <sup>131</sup>, or to individualize training exercises to ADHD patients' pre-existing executive deficits <sup>132</sup> also have not held up against placebo control. Most reviewers of this literature have concluded WM training still holds considerable promise in ADHD <sup>108, 109, 112, 113, 115, 117, 133-138</sup>. But they also make it clear new ideas are needed for how to modify training to have stronger and more reliable benefits for ADHD symptoms. We believe meaningful ADHD clinical improvement will require not only an entirely new cognitive training focus, but also a neuroscience-informed research formulation that identifies brain-based training targets that have been empirically shown to predict ADHD symptom expression.

Executive Working Memory This proposal builds on converging theory and evidence that 'executive working memory' (EWM) likely represents a better context for ADHD WM training than WM storage capacity, with highly specific brain-based training targets of clear relevance to ADHD. EWM describes cognitive operations that account for what Baddelev's seminal WM theory described as the 'central executive' – a system that controls information flow within WM. Although early WM studies tended to conceptualize WM's central executive as a single construct, neuroscience evidence suggests that instead there likely are a small number of behaviorally dissociable basic EWM operations supported by partially overlapping brain systems. Bledowski et al. <sup>139</sup> has proposed some of these EWM operations promote *flexibility* of selective attention to WM contents (e.g., measured by tasks that require attention Shifting among information held briefly in WM or Updating WM content with new information). Others lend stability to WM representations (e.g., Filtering any extraneous distracting information during WM maintenance, or Suppression of proactive interference from uninformative information during retrieval of information from WM) 140. These attention-based EWM basic operations emerge directly from Cowan's 54, Oberauer's 141, and Engle's 142, 143 current theories about WM's central executive and reflect a basic, well-supported dichotomy between maintenance vs. disengagement via selective attention processes 144. Each of these EWM operations seem to be suitable candidates for cognitive training exercises. To justify combining them all into a unified EWM training intervention, we examined their relationship to each other in N=160 adults who completed online EWM tasks on Amazon's mTurk internet worker platform 145, 146, and whose data met rigorous sampling and data quality control criteria 147-149. These participants completed the same verbal and nonverbal versions of the EWM Updating, Shifting and Distractor Filtering/ Suppression tasks we propose to use in this project (See Approach). Confirmatory factor analyses of EWM task accuracy found acceptable model fit for both a 1-factor model where all EWM accuracy scores contributed to a single latent EWM construct (i.e., GFI=.947, RMSEA=0.072), and a 4-factor model showing each type of EWM ability had unique variance (GFI=.971, RMSEA=.049, and a non-significant CMIN test p=.155). This combination of shared and unique variance supports that they all fit underneath an umbrella EWM construct, but also that none of the EWM operations could be considered redundant. As such, all seem to be viable candidates for EWM training exercises.

Neurobiological Basis of EWM EWM operations have been extensively studied with fMRI 151-174. Meta-analysis of EWM-specific fMRI studies 140 (Fig. 1) find EWM operations overlap with a core frontoparietal WM representation network for information encoding, storage and retrieval (Fig. 2) found by meta-analysis of literally hundreds of fMRI studies, but engage a more extensive set of brain regions throughout lateral/medial PFC and parietal cortices. Current 'state representation' WM neural models describe how the core WM network is integrated with these EWM-linked regions via selective attention mechanisms that activate and integrate information processed in distal regions. This engages information in an active form that can be manipulated and used to guide behavior (sometimes termed 'primary memory' 112, 175-177). Within this state representation



theoretical context, the so-called 'working' parts of WM are simply these various specific attention-based EWM processes – *Shifting*, *Updating*, *Filtering*, and *Suppression*. D'Esposito and Postle <sup>178</sup> recently gave a cogent summary of the considerable neurobiological evidence for how WM arises from such attention-related network connectivity changes during EWM task performance. That is, functionally heterogeneous <sup>179-182</sup>, hierarchically-

organized <sup>183-185</sup> prefrontal cortex (PFC) regions engage sustained activation <sup>186-188</sup> during WM that biases activity in other PFC brain regions or other parts of the brain in a 'top-down' way <sup>189-191</sup> via synchronized activation <sup>192, 193</sup> to support WM state representations for information manipulation. Two brain regions seem to be particularly important for these EWM operations – caudal superior frontal sulcus (SFS) linked to feature prioritization

within WM 140, and a mid-lateral PFC region of the inferior frontal junction (mid-latPFC), immediately below and posterior to BA 9/46 linked to selecting among competing contexts or rules. Meta-analysis shows that SFS and mid-latPFC are engaged for all EWM operations, possibly because they are key nodes in 'where' and 'what' WM information selection systems <sup>140</sup>. We demonstrated the importance of these regions in pilot Dynamic Causal Modeling (DCM) 194, 195 analyses of EWM fMRI task data that characterized causal relationships among EWM task-engaged brain regions (Fig. 3). While extensive details are not necessary to illustrate the key point, SFS and mid-latPFC exert direct excitatory causal influences on other prefrontal and posterior brain regions engaged for EWM. Those influences also are strongly correlated with behavioral accuracy. The position of SFS and mid-



Fig. 3A: Dynamic Causal Modeling results in n=15 adults during EWM Updating. GREEN dashed lines show excitatory intrinsic causal influences; RED inhibitory influences (Cohen's d > .50). Fig. 3B: Specific DCM matrix B modulatory connections that are + or - correlated r > .35 ('medium' effect size) with Updating task % accuracy. 88% of connections involved mid-latPFC (IFJa) or SFS (55b) parcels.

latPFC near the top of EWM network hierarchy and their role as ubiquitously-engaged information processing nodes for many types of EWM operations make them promising EWM training target candidates.

Support for EWM as a Training Focus in ADHD Here, we review neuropsychological and neuroimaging evidence that supports EWM is meaningful in ADHD and that SFS and mid-latPFC EWM-related brain regions have a plausible relationship to symptom expression. First, *meta-analysis shows EWM deficits are by far the strongest WM deficits in ADHD*. Meta-analytic statistical comparison finds they EWM deficits are significantly stronger than WM storage <sup>72</sup> in ADHD (p<.037 for verbal; p<.022 nonverbal). Moreover, if one re-arranges the 64 ADHD deficits Hedge's g effect sizes from this meta-analysis g, the simplest short-term storage tasks' have an average g=0.54 ("medium" deficit), while low executive demands like reversing information before recall g=0.72 ("large"). The greatest ADHD effect size impairments (average g=1.13; very "large") were seen for very high executive WM demands, such as switching attention among concurrently held information sets, etc. This EWM effect size also is notably larger than any other cognitive impairment linked to ADHD (e.g., response inhibition, set shifting, timing, etc. g=1.13 (so perhaps one reason prior ADHD WM storage training trials have failed to benefit clinical symptoms is they have not targeted the most-impaired WM abilities that have the greatest likelihood of being related to the brain dysfunction central to ADHD.

Second, <u>fMRI EWM studies offer clear treatment targets because they reliably converge on specific ADHD brain abnormalities</u>. Functional MRI study reviews and meta-analyses fail to precisely localize abnormalities in ADHD brain regions activated by simple WM information storage tasks <sup>76, 199, 200</sup>. Close examination shows no two ADHD fMRI WM storage studies <sup>103-106</sup> have localized ADHD abnormality to exactly the same brain region. In contrast, fMRI studies consistently find evidence for ADHD dysfunction in brain regions specialized for EWM operations <sup>201-210</sup>. For instance in McCarthy et al.'s meta-analysis <sup>211</sup> of 4 fMRI studies that used an N-Back WM task (which engages EWM operations on each trial – *Shifting*,



Fig. 4. Comparison of non-ADHD (n=5) > ADHD (n=5) executive WM fMRI Cohen's d effect size maps for activation and connectivity. Maps thresholded at d > 0.50 ("medium" effects).

*Updating*, and *Suppression* <sup>212</sup>), ADHD hypofunction was reliably found in the same bilateral SFS and medial PFC regions. To date, only 1 ADHD fMRI study has attempted to localize neural dysfunction to a specific, isolated EWM operation (i.e., distractor filtering <sup>106</sup>). It also found findings consistent with our conceptual model – lower ADHD intra-PFC functional connectivity, and blunted WM load-dependent activity increases in left ventrolateral PFC, right insula and right medial PFC. Again, these are mostly regions implicated in EWM instead of the 'core' WM representation network. Fig. 4 shows pilot study results that bolster confidence that impaired ADHD

activation in SFS, mid-latPFC and other EWM-linked brain regions is found during all EWM operations we propose for the new intervention. (Note, this pilot study used fMRI analysis methods and a cortical atlas developed by the Human Connectome Project (HCP) that refers to discrete brain regions as HCP atlas 'parcels'.) During WM *Updating*, ADHD had less activity in bilateral dlPFC parcel p9-46v and parcel PF (in the supramarginal gyrus; SMG). ADHD had lower activation to parcel AAIC (insula) to recall probes on the WM *Suppression* condition – an effect made more prominent in the presence of proactive interference. For *Distractor Filtering*, ADHD had less activation of parcel 7PL (superior parietal lobule) and parcels in both dorsal and ventral regions of bilateral PFC. Several bilateral dACC parcels were hypofunctional during *Distractor Filtering* and *Updating*. ADHD functional connectivity estimated by graph theory-based methods <sup>213-216</sup> was weaker connectivity in parcel 55b (caudal SFS) in the *Suppression* task, parcel PGi (SMG) for *Updating*, and tasks in SPL parcels 7PC and 7AL for *Filtering*.

Third, if the ultimate goal of ADHD WM training research is to reduce ADHD symptoms, we suggest the most suitable brain treatment targets are those with a convincing association with ADHD symptom expression. Very often, only a subset of brain abnormalities found to be abnormal within a given psychiatric diagnostic phenotype has a direct association with the severity that disorder's symptom expression. In the largest study of ADHD brain structure abnormalities ever undertaken (N=2.246 ADHD patients), the ENIGMA consortium found throughout all cortex that only a superior frontal gyrus region (r=-0.19, p=0.01) (i.e., encompassing our proposed SFS target) and rostral cingulate (r=-0.18, p=0.03) surface area measurements were associated with ADHD Hyperactive/Impulsive symptom severity. Surprisingly few published ADHD fMRI studies examined brain activity correlations with symptom severity in post hoc analyses (only 6 of >6 dozen reports we reviewed). Nevertheless, there is piecemeal evidence that links ADHD symptom severity to lateral PFC. One study found a correlation between symptom severity and right lateral PFC activation during WM for emotional stimuli <sup>207</sup>. Another found a link between lower ADHD symptoms and methylphenidate-induced normalization of Stroop task-elicited left dIPFC activity 217. Another type of evidence for a link between WM change and ADHD symptom change recently was found in a prospective study that showed normative improvements in ADHD patients' WM ability from childhood to early adolescence directly predicted lower ADHD symptoms in patients <sup>218</sup>. This was a specific relationship, as similar developmental gains in



corrected). Data from 103.

response inhibition and sustained attention ability did not predict symptom levels. All these indications are suggestive, but admittedly limited. However, even stronger evidence exists linking ADHD symptom reductions to activity changes in our specific proposed EWM-related brain targets. In our recent R21HD061915 study, we examined the effect of 5 weeks of Cogmed™ WM storage training on ADHD adolescent brain activation elicited by a WM fMRI probe <sup>103</sup>. After training, ADHD PFC activity elicited during WM storage improved to non-impaired levels (Fig. 5). However, those WM storage-related neural gains did not predict clinical improvement. Instead, when meaningful clinical improvement was seen (in 61% of the ADHD sample), symptom reductions correlated with increased activity in brain regions known to be functionally specialized for EWM <sup>139</sup> (e.g., bilateral SFS, ventrolateral PFC, pre-SMA, and IPL/SMG and SPL parietal lobe regions). These findings not only provide clues as to why WM storage training fails to reduce ADHD symptoms (i.e., it targets the wrong brain regions), it offers a strong indication that EWM brain region change underlies ADHD symptom remission. Because Cogmed™ exercises have minor executive demands, our observations likely resulted from an unintended, coincidental strengthening of EWM-related neural circuits despite Cogmed™ targeting of WM

storage. Interestingly, our findings showed only the caudal SFS gains correlated with improvements in *both* Hyperactive/Impulsive and Inattentive symptoms, suggesting it might have relatively greater therapeutic potential than other regions.

Finally, we conducted a proof-of-concept pilot study to show *EWM training alters ADHD activity and functional connectivity in the proposed brain treatment targets. N*=7 ADHD-diagnosed adolescents drilled on all EWM operations in exercises over a brief, 2-week course of practice (6 sessions). Fig. 6 depicts widespread increased brain functional connectivity to the right SFS parcel in different EWM task contexts after EWM practice. Both 'large' and 'very large' effect size connectivity increases were seen, within 'core' WM and EWM-specialized



Fig. 6. ADHD brain regions that increased their functional connectivity with right Superior Frontal Sulcus (SFS) HCP 'seed' parcel [55b] (outlined in turquoise) after 6 EWM training sessions. Maps are thresholded at d > 1.0 ('large' effect sizes).

regions, as well as with other brain regions. Interestingly, different connectivity changes were seen when brain function was elicited by different EWM tasks, consistent with WM state representation theories that the key SFS and mid-latPFC regions will dynamically reconfigure their connectivity strength for different EWM demands. Therefore, we are likely to have the most widespread effect on EWM neural network function if we include all 4 different EWM operations as training exercises. Although this is strong evidence of these regions' malleability and responsiveness to EWM practice, the next step of this research is to give patients a typical course of WM training (e.g., 20-25 sessions over 5 weeks) to assess the extent of brain target engagement with fMRI analyses of activation and network connectivity. In this pilot, behavioral gains were not expected because participants only performed rote practice. Actual EWM training will adaptively increase task difficulty and include intervention design elements that ensure engagement and motivation. These are essential ingredients generally believed necessary to alter behavioral performance <sup>43</sup>.

Synthesis and Potential Impact There generally is increasing enthusiasm and optimism for using cognitive training to treat psychiatric disorders as more and more studies discover its principles of application, and document its ability to re-sculpt brain networks through experience-dependent neuroplasticity <sup>219</sup>. Although the basic premise underlying some sort of WM training in ADHD still seems sound, a WM storage training behavioral target has been proven ineffective. Broadly speaking, it makes sense that any link between WM and ADHDrelated behavioral impairment is likely to be more greatly related to patients' ability to effectively use the information represented in WM in the service of cognition and behavioral control instead of merely how much information can be temporarily held in WM. Guided by a careful synthesis of neuroscience evidence from the past decade, this proposal argues for new EWM-focused exercises as a vehicle for modifying specific new brainbased targets. To recap, we conceptualize EWM impairments as the behavioral manifestation of a dimensional, RDoC-like <sup>220-224</sup> neurobiological abnormality in patients diagnosed with ADHD. Although not all ADHD patients show every cognitive impairment that has been linked to the diagnostic phenotype 64, 77, 225-228, EWM tests have the strongest effect size of any cognitive impairment in ADHD. This suggests EWM impairments are more important, or perhaps expressed in a greater proportion of ADHD patients than WM storage or other executive deficits. Cognitive neuroscience neuroimaging studies point to SFS and mid-latPFC as ubiquitously important for all EWM operations; they direct the dynamic reconfiguration of EWM neural network function when accessing or protecting information held in mind to direct behavior that predict EWM task accuracy. Clinical neuroscience studies also show these regions have abnormal activation in ADHD during EWM task performance and are linked to ADHD symptom expression. As such, these two regions represent potential intervention targets whose engagement likely have a stronger potential to produce ADHD symptom severity or functional level improvements that have been so elusive in prior WM storage training research (e.g., Cogmed<sup>TM</sup>). We contend brain-based training targets ultimately will prove better than behavioral performance-based targets because they are more proximal to putative disease mechanism. In this context, EWM behavioral change remains an important focus of cognitive training interventions, but primarily for interpretive reasons (i.e., to ensure training exercises have the intended effect). Furthermore, our consideration of EWM brain region inter-connectivity to evaluate target engagement is consistent with the most recent ADHD neurobiological models of the disorder stemming from neural network connectivity abnormalities <sup>229-237</sup>. It also is noteworthy that success here is potentially relevant for other disorders whose putative etiology is linked to WM (e.g., schizophrenia and bipolar illness 238<sup>240</sup>, TBI <sup>241</sup>, MS <sup>242</sup>, stroke <sup>243</sup>). A successful target engagement demonstration here might open new therapeutic avenues for any disorder that shares diagnostically cross-cutting abnormalities in EWM abilities.

The R61/R33 phased grant mechanism for efficient experimental therapeutics development is ideal for the current stage of this research. The obvious next step is to repackage the EWM probes used in prior neuroscience research into a multi-week, intensive drilling format commonly used to maximize participant engagement and to continually challenge EWM ability. Two carefully designed clinical trials will let us determine if the SFS and midlatPFC targets are indeed engaged by EWM training, to replicate findings, and assess if target engagement has clinical relevance – all necessary to support future clinical efficacy testing. There should be optimism for success because a small handful of EWM training trials already have shown some success in both ADHD 244, 245 and non-ADHD samples 92, 136, 246-249, at least at the behavioral performance level. Those studies trained comparable EWM operations to what we propose to study here. But they typically did not ensure training on all possible EWM operations linked to the proposed SFS/mid-latPFC brain targets. Moreover, we focus here on both brain and behavioral levels. The R33 will examine a larger replication sample. It will test 'near-transfer' generalization, and consider training delivery and patient characteristics as potential outcome moderators (e.g., pre-existing WM impairments vs. strengths, sex, age, ADHD subtype, etc.). These analyses will ensure target engagement evidence meets all theoretical expectations and is robust to the likeliest potential confounds. By the end of this R61/R33 project, we either will know to abandon this proposed new line of inquiry, or we will be positioned to conduct one of several possible 'next step' studies. Ideally, we expect to be ready to propose a well-informed preliminary clinical efficacy trial. Alternatively, we may learn we need to optimize the intervention delivery based upon the results of some proposed R61/R33 supplemental analyses that will determine if target engagement is moderated by the pace of EWM gains, exposure to training (i.e., 'dose'), or patient characteristics.

Innovation The primary study proposal innovations are the new EWM treatment target and its primary focus on neurobiological targets presumably closer to ADHD etiology. Despite strongly converging evidence, none of these EWM operations have been explored in depth in ADHD at the brain level, either in ADHD itself or within a cognitive training context. Another important novel feature is our successfully-piloted remotely-supervised 'at home' EWM training that effectively substitutes for in-person appointments. Not only should this delivery approach greatly enhance protocol adherence and retention, it provides a potentially paradigm-shifting option for a way to deliver personalized cognitive training that should prove to be more practical for typical families in future efficacy trials. There also are many advantageous clinical trial design elements and analyses we describe in the Approach that were not used in most prior ADHD WM training trials. These should overcome common clinical trial pitfalls to help ensure the most definitive possible answers to our target engagement hypotheses.

### APPROACH - Methodology in the R33 Project Phase

**Participants** ADHD participants in the R33 (n=90) trial will be representative of adolescents with a primary diagnosis of DSM 5 ADHD who have common minor secondary psychopathology (see the Eligibility Criteria section). The R33 also will recruit n=40 demographically-equivalent non-ADHD participants for a useful comparison of ADHD EWM performance and brain function against a typical normative sample. We focus on adolescent ADHD rather than children in part to avoid pre-pubertal neural differences and to continue our prior ADHD fMRI research (all of which focuses on teens). But also, adolescence represents an ideal developmental period for neuroplasticity-based interventions. It has been well-established that post-pubertal neural system changes mostly involve experience-dependent refinements to a largely-established 'adult-like' brain organization (see our recent adolescent network connectivity review <sup>250</sup>). We are experienced from nearly a dozen current and recent Ro1s with large N recruitment for fMRI studies of adolescents. As in our recent R21HD061915 and Ro1MHo80956 ADHD fMRI studies, ADHD participants will be recruited from both clinical and community resources. ADHD is ~4 times more common in boys <sup>251</sup>, but we will over-sample ADHD females to assess sex effects on outcome, as per NOT-OD-15-102 (> 1/3 will be female). A Note on ADHD Medications: All 'in person' visits for ADHD fMRI/neurocognitive evaluations will require a 24-hour medication washout if patient symptoms are managed with typical, short half-life psychostimulants. This is a common, widely-accepted research practice to ensure test results cannot be attributed to the temporary, palliative effects of those drugs on the brain on assessment days (see Eligibility Criteria section for detailed discussion of the issues involved and list of permitted medications).

Clinical **Assessment** This evaluation will fully assess all the study exclusion criteria and quantify symptom severity ADHD functional ability. Table 1 lists evaluation instruments, noting when multiple respondents will provide subjective ratings. All measures are validated for adolescents. As per K-SADS-5 guidelines, collateral parent interview will inform diagnosis decisions. Diagnostic interviews will be performed by clinically-trained

| Table 1. Clinical Assessment (R61/R33) | | |
|---|---|---|
| Task Name | Domain | Min |
| K-SADS-5 <sup>252</sup> | DSM Axis I diagnosis | 30-120 |
| Child Behavior Checklist (CBCL) <sup>253</sup> | Psychiatric/problem behavior | 10 |
| Conners 3 (P/S) <sup>254</sup> | ADHD symptom severity | 20 |
| * Weiss Func Impair Rating Scale (P/S) <sup>255</sup> | Psychosocial function | 5 |
| * Inven. of Parent and Peer Attach. (P/S) <sup>256</sup> | Social relationship quality | 10 |
| * Wide Range Achievement Test-5 | Academic Achievement | 45 |
| Beck Depression Inventory II <sup>257</sup> | Depression severity | 5 |
| Multidimen. Anxiety Disorder Scale 2 <sup>258</sup> | Anxiety | 5 |
| Olin Health Care Questionnaire | Health and substance use | 10 |
| Adol Alcohol/Drug Involv. Scale (AADIS) <sup>259</sup> | Alcohol/Drug involvement | 5 |
| Fagerstrom (FTND) <sup>260</sup> | Smoking status/nicotine use | 1 |
| Petersen Physical Develop. Scale <sup>261</sup> | Pubertal status | 5 |
| * Clinical severity measures to assess functional impairment; P – Parent, S – Self | | |

postdoctoral staff supervised in a weekly diagnosis consensus meeting by PI Stevens (a licensed clinical psychologist with >16 years' experience supervising K-SADS interviews for NIH-funded studies). Staff interviewing training will include 10 "modeled" interviews, direct observation of the first 10 interviews, and quarterly review of all interview videotapes by other clinically-trained research staff to control for assessment 'drift'. We also will assess participants' age, race/ethnicity, education level, handedness <sup>262</sup>, and socioeconomic status <sup>263</sup>. Parents will detail family psychiatric history <sup>264</sup> and confirm child's medical history. These clinical evaluations usually last between 2 - 3 hours.

**Neurocognitive Assessment** Cognitive testing will exclude WASI FS IQ <sup>271</sup> <80. It also will detail common WM processes, assess EWM tests of 'near transfer' to test the generalizability of EWM training outside of trained tasks, and test 'far transfer' of training effects to other abilities often impaired in ADHD. Table 2 lists tests along with their test-retest reliability. Cognitive testing will require ~2 hours. Co-I Dr. Hawkins will supervise staff training and cognitive testing procedures throughout the project.

**MRI** Assessment Overview MRI data will be collected using a Siemens 3T Skyra. Subjects will wear hospital 'scrubs' to minimize the chance of introducing metal into the MRI. They will provide a urine sample before MRI to test for drug metabolites, and pregnancy

| Table 2. Cognitive Tests (R61/R33) | | | |
|---------------------------------------|-----|-------------|-----|
| Domain/Task Name | Ref | Reliability | Min |
| Working Memory Capacity | | | |
| WISC-IV Letter-Number Sequencing | 265 | .90 | 15 |
| WISC-IV (Integrated) Spatial Span | 265 | .7981 | 5 |
| WISC-IV Digit Span | 265 | .8083 | 5 |
| EWM 'Near Transfer' Tests | | | |
| Shifting – Refresh/Repeat Task | 156 | n/a | 12 |
| Updating – Spatial Updating Task | 266 | n/a | 14 |
| Filtering – Attend-Ignore Task | 172 | n/a | 4 |
| Suppression - Intr. Resistance Task | 160 | n/a | 12 |
| Executive/Other Abilities | | | |
| CPT-II Omissions (Sustain. Attention) | 267 | .84 | 15 |
| CPT-II Commissions (Resp. Inhib.) | 267 | .65 | - |
| CogState Detection (Process Speed) | 268 | .92 | 2 |
| CogState Set Shifting Task (Shifting) | 268 | n/a | 5 |
| Temporal Estimation Task (Timing) | 269 | n/a | 6 |
| Stroop Color/Word (Cog Control) | 270 | 0.97 | 6 |

in females. Positive drug results could defer MR data collection and will be noted for *post hoc* analyses. Caffeine/nicotine intake and cigarette smoking will be as normal to prevent acute withdrawal effects on brain activity, but restricted to >1 hour prior to MRI to avoid well-documented neural effects of recent use.

**fMRI Paradigms** There are two important differences between the fMRI tasks that will assess EWM ability before and after training and the EWM training exercises. First, 4 separate tasks will be used during training to isolate each EWM operation, whereas fMRI uses 3 because WM *Distractor Filtering* and WM *Suppression* can be efficiently combined into a single paradigm. WM *Updating* and WM *Shifting* cannot be evaluated by fMRI simultaneously because each operates differently on the stimuli set held in WM. In contrast, EWM stability operations can be assessed in using the same trials because the EWM operations take place after WM short-term maintenance <sup>272</sup>. By combining them for fMRI, we lessen the fMRI scanning time burden. Second, to avoid stimulus familiarity confounds the fMRI tasks will use stimuli sets never seen during EWM training (different counter-balanced sets between pre-/post-training MRI scans). Because SFS and mid-latPFC engagement has proven by meta-analysis to be largely domain-general <sup>140</sup>, we include both verbal and nonverbal versions of each task with the expectation they will be collapsed for stable measurements. The

visuospatial versions will use fractal images that are not easily encoded verbally. All were constructed with adequate delays for WM maintenance, but not so long to raise concerns over different WM decay times or possible use of undirected rehearsal strategies. Because it is crucial we avoid exceeding typical WM storage span (which could result in our study testing WM storage capacity more than EWM), no exercise uses more than 4 stimuli at a time (i.e., this is the well-replicated limit of the primary memory span <sup>54</sup>). Task visual layout and pacing are similar so any cross-task differences can be confidently attributed to the EWM operations themselves.

<u>WM Updating</u> This task measures replacement of items in WM. It is based upon Murty et al. <sup>273</sup>, simplified to 2 conditions. Each trial begins with 4 stimuli presented for 4 sec, followed by 2 to 4 successive presentations (2 sec each) of an asterisk as placeholder or a new stimulus in each position (Fig. 7). For asterisks, participants are instructed to retain the previously viewed stimulus in WM, but to update the contents of WM for any new stimulus. During a final 3 sec response phase, participants indicate if the presented stimuli match the contents of WM (half the probes are correct/half incorrect). For fMRI, the primary contrast of interest is Updating > Maintenance. Each of two fMRI runs (verbal or visuospatial) has 20 Maintenance and 20 Updating trials. Each run=11:39 min (23:18 total).

<u>WM Shifting</u> This task measures the ability to refocus selective attention to different stimuli held concurrently in WM without altering WM contents. Each trial (Fig. 8) begins with 4 stimuli (verbal or visuospatial) for 4 sec, then a 6 sec delay with no stimuli. In a 4 sec probe phase, one location is highlighted and subjects are cued to respond to different Yes/No questions about item content (i.e., randomly chosen to ensure participants do not just encode answers instead of stimuli). For verbal – "Alive?" vs. "3 Letters?" For visuospatial – "Color?" vs. "Fills Screen?"). For Control trials, subjects are

Memory Set (4 sec) MAINTENANCE UPDATING (6 sec) (3 sec) "Correct or Incorrect?" Fig 7. WM Updating Task trial. Memory Set Delay **Probe** ROPE PIG KITE (4 sec) Fig 8. WM Shifting Task Trial

prompted to hit a randomly-chosen button. For fMRI, the contrast of most interest is Shift > Control. Each of two fMRI runs (verbal or visuospatial) has 12 Control and 12 Shift trials. Each run=7:10 min (14:20 total).

<u>WM Distractor Filtering/Interference Suppression</u> This task assesses brain function engaged to a) suppress/inhibit irrelevant, distractor information from WM and b) suppress proactive interference during WM retrieval <sup>272</sup>. Participants are asked to retain a 4-item memory set in WM (Fig. 9). For the verbal task, two stimuli are shown in red, two blue. Our visuospatial version has a comparable format, except instructions are to retain the two top or bottom stimuli.



After a PreCue retention-interval, a 2 sec Cue instructs participants to retain in WM only items of that color (i.e., 50% red or 50% blue) throughout a PostCue WM retention-interval. A probe word requires an affirmative dominant-hand response if it matches either of the items retained in WM (e.g., POOL and TILL). On 50% of trials the probe matches one of the items that should be in WM (Valid probes), on 25% the probe matches one of the items that should have been inhibited from WM (Lure probes), and on the remaining 25% of the trials the probe does not match any WM items (Control). For fMRI, the contrasts of interest for this study are PreCue > PostCue (efficacy of suppression) and Lure > Control probe (resolution of proactive interference). Each fMRI run=5:28 min (21:52 total).

**Stimulus Delivery/Response Recording** E-Prime (Psychology Software Tools, Inc.) will implement fMRI tasks. Stimuli will be projected via a 3200 ANSI lumens system onto a screen behind the patients head in MRI. Participants view this screen using a mirror on the head coil. An MR-compatible 5-button fiber optic response device (Current Designs, Inc.) will acquire behavioral responses. Each fMRI task is programmed to track accuracy and RT for conditions of interest for offline analysis. Participants communicate with staff during MRI using an MR-compatible auditory sound system delivered by 30 dB sound-attenuating headphones.

**MRI Sequences** *fMRI* gradient EPI (TR/TE 900/35 msec, flip 60°, multi-band AF=7). *Fieldmaps* (TR/TE 8400/62 msec, flip 80°, AF=1, 0:25 min, run twice with reversed A>>P phase encoding) (EPI/fieldmap

sequences have 2.1 mm isotropic voxels, 70 interleaved slices, 228 mm FOV). <u>T1-weighted</u> (3D MPRAGE, TR/TE/TI=2400/2.07/1000 msec, flip 8°, FOV=256×256mm, 0.8 mm isotropic vox; 7:02 min). <u>T2-weighted</u> (TR/TE=3200/565, FOV=256x256, 0.8 mm isotropic vox; 6:45 min). Images will be Radiologist-assessed to be free of macroscopic pathology. Daily MR stability/QA will ensure equal scan quality throughout the project.

HCP Pipeline MRI Processing We have experience with Human Connectome Project (HCP) <sup>274</sup> preprocessing pipelines <sup>275</sup> from several prior and ongoing large Ro1 MRI studies. They provide highly-accurate, structural image-guided brain atlas normalization for fMRI data. T1/T2 images will be ACPC-oriented, brain extracted, B<sub>o</sub> inhomogeneity-corrected, mutually co-registered, distortion fieldmap-corrected, and finally MNI152 atlas-registered using FSL FLIRT+nonlinear FNIRT algorithms <sup>276</sup>. FreeSurfer-based <sup>277</sup> registration, skull-stripping, and pial extraction on 1mm downsampled T1/T2 data will create structural volume/cortical ribbon files. After fMRI EPI data is motion-corrected, it will be registered to FreeSurfer output, resampled to atlas space, intensity normalized, smoothed (cortical ribbon surface mapping data @2mm FWHM), and written as timeseries in CIFTI format for analysis. All fMRI analyses will examine brain regions localized to the cortical subdivisions identified by the recently released HCP multimodal-derived map of 180 cortical parcels <sup>278</sup>. We emphasize this point, as this atlas represents the highest-resolution cortical atlas to date, including 97 new regions. It divides conventionally-recognized structures into numerous sub-regions defined by uniquely demarcated boundaries constructed using each brain's functional connectivity and myeloarchitecture. We also will use a recently-developed sub-cortical/cerebellar map that reveals 358 highly-organized parcels that align with these new cortical regions <sup>279</sup>. Together, these atlases represent the cutting-edge in brain localization.

MRI and Head Motion Total MRI session time is 1h 10 min, of which 50 min involves fMRI data collection. Although this scan duration can be challenging for adolescents who are prone to fidget (especially unmedicated ADHD participants), we have ample experience scanning ADHD teens (Ro1MHo8o956, R21HDo61915, K23MHo7o036) and non-ADHD teens for these scan lengths. A mock scanner will acclimate subjects. Framewise Integrated Real-Time MRI Monitoring (FIRMM; <a href="https://www.firmm.io">www.firmm.io</a> <sup>280</sup>) will prompt staff to discontinue obviously unusable scans (i.e., data with movement >1 2.1 mm voxel); these will be replaced with parallel task versions in the same session. This will be more time/cost-efficient than a 2<sup>nd</sup> scan. If needed, substitute scans at a proximal session will be done to avoid discarding an entire dataset. Minor head motion or sharp spikes will be addressed using ICA-FIX <sup>281, 282</sup>, which isolates/de-noises such signal artifacts and regresses linearly-detrended motion parameters from the HCP-processed timeseries. We have learned in 15+ years of pediatric fMRI experience >90% of adolescent non-ADHD and >80% of ADHD fMRI data meets QC criteria, while roughly 10% of ADHD ultimately can be replaced by a second scan session with careful participant re-training.

**Conventional fMRI Analyses** Single-subject activation will be quantified with FSL FEAT with FMRIB's Improved Linear Model, using geodesic Gaussian algorithms to estimate autocorrelation and smooth surface-based fMRI data. Explanatory Variables (EVs) will use a double-gamma HRF convolution to translate event onsets in conditions-of-interest into regressors to be fit to the BOLD timeseries. EV contrasts (against other conditions) will create activation maps. Task performance will be considered by 1) separately modeling correct vs. incorrect events, then collapsing across them if SFS/mid-latPFC measurements are unaffected by accuracy, and 2) examining the effect of accuracy for *post hoc* analyses at the group-level.

Functional Connectivity Analyses Graph theory (GT) offers a diverse variety of useful and informative network metrics. In GT, networks are mathematical representations of real-world complex systems. GT metrics parameterize these systems to describe relationships among fMRI-measured region activity profiles 283, 284. GT metrics range from those that simply quantify how integrated a single brain region is with others in a network or sub-network, to others that capture more complex properties of network structure, integration, segregation, or resilience to insult 215. Although it is possible to examine thousands of connections among SFS, mid-latPC and other relevant brain network regions. GT also can focus hypothesis-testing on individual brain regions to reduce multiple comparisons demands. Our primary functional connectivity metric will be 'weighted-degree,' which quantifies the number of edges (connections) to a any network node of interest, weighted by their association strength. In this way, we will have a single value per participant for SFS and mid-latPFC parcels that represents nodal functional connectivity strength. When preparing data, we will follow detailed published recommendations to mitigate any head motion signal artifacts <sup>285, 286</sup> on fMRI timeseries data. Because ICA-FIX already will have been applied and motion parameters regressed from the data from HCP processing, we additionally will regress white matter, CSF and global signal from the data, then apply a 0.8 Hz low-pass filter. The residualized timeseries will use partial correlation to form adjacency matrices <sup>287</sup>. Un-thresholded, full adjacency matrices will avoid the arbitrariness of threshold selection and loss of information when binarizing connections.

**EWM Training Trial Methodology Considerations** Although the primary purpose of the R61 and R33 trials is a to assess target engagement, not clinical efficacy, the major criticisms of prior ADHD WM training efficacy trials noted in reviews of the available literature <sup>109, 112, 113, 115, 134-137</sup> provide design considerations that are germane to any cognitive training trial. These issues are summarized in Table 1, along with our innovations to avoid the same limitations to enhance this project's methodological rigor and potential reproducibility.

| Table 3. Methodological Criticisms of Previous WM Training Clinical Trial Design or Interpretation | |
|---|---|
| Issue | Solution |
| Active placebos in RCTs also can produce clinical improvement, | Use a carefully-chosen placebo arm, and supplement with other |
| possibly undermining clear understanding of WM training efficacy | methods for ensuring any gains after EWM training are valid |
| RCTs do not examine how treatment compliance affects outcome | CACE analysis of the effect of compliance on WM outcome metrics |
| EWM test performance at trial outcome might be contaminated by practice effects | Ensure stimuli used for training are not used for pre- and post- |
| | training fMRI assessment; for all WM neuropsych tests used for |
| | assessment, choose those with reliable parallel forms |
| Near- and far-transfer inconsistently evaluated | Include commonly-used tests for comparability across studies |
| Not all previous studies evaluated psychiatric comorbidity (e.g., | Conduct full diagnostic interview and assess possible academic |
| CD/ODD), ADHD DSM-IV clinical subtype, or LD | disparity with IQ; evaluate outcome moderation effects statistically |
| The medication status of ADHD participants has been inconsistent | Limit to unmedicated ADHD and those on stable, short-acting |
| and often un-evaluated across studies | psychostimulants; use 24 hour "washout"; assess moderator effect |
| Not clear to what extent age influences one's ability to benefit from | Avoid pre-pubertal children to circumvent major developmental |
| executive WM training; possible pubertal confounds | confounds; examine age (or time since puberty onset) moderation |
| Previous studies typically ignored any effects that individual | We will randomly assign participants to active/placebo treatment |
| differences in pre-training WM ability might have on outcome | and examine the role of pre-training EWM ability on outcome |

**Placebo Condition** The strongest criticisms of prior ADHD WM training RCTs are the absence of placebo control, as results could be driven by expectancy effects. Although neural and neurocognitive measures of target engagement that are the focus of this project are less vulnerable to expectancy, we chose to add a placebo training group to both R61 and R33 for methodological rigor and to enhance the certainty of causality inferences. Choice of placebo for WM training trials is challenging because some previously-used WM 'active placebos' have changed brain function <sup>288</sup>. We will use Mahjong and Bejeweled tile games for the placebo condition. These deliver an equivalent 'training time' exposure, are compatible with remote monitoring, the game elements can be presented as a feasible treatment to preserve the blind, and we provide the same coaching experience. We only will use these tile games for placebo exercises as they have low EWM demands <sup>196, 197</sup>.

Executive WM Training Sessions Each ~50 min EWM training session will include sixteen 3 min EWM exercises (counter-balancing the order of EWM task types and verbal vs. nonverbal versions). To avoid stimulus familiarity effects, the stimulus set for all exercises will be unique each training day, drawn randomly from a large pool. Importantly, EWM training task difficulty will be adaptively increased across the 5 weeks of training based on session-to-session performance. Day 1 EWM training will begin with relatively easy 2-item memory sets. These will quickly ramp up to 4-item stimuli sets across the first 2-3 sessions as each participant attains 80% accuracy for each 3 min exercise. After this familiarization/confidence-building period across the 5 Week 1 sessions, EWM task difficulty manipulations will begin using an adaptive staircase design. Each EWM exercise will manipulate difficulty in different ways. For WM *Updating*, the number of updates per trial will increase from 1 to 4. If a participant achieves proficiency when challenged by 4 WM updates, the speed of each update will be shortened by 100 msec until behavioral gains plateau or a minimum of a 1 sec response window. For WM Shifting, the number of shifts per trial will be increased from 1-4, then duration of each response window successfully shortened by 100 msec. For WM Distractor Filtering, the number of possible colors used for directed forgetting will be increased from 2 to 4, then response window shortened by 100 msec. For WM Suppression, more proactive interference probes will be given at once (from 1 to a max of 4), then 100 msec response window will decreases once consistent optimal performance on 4 probes is attained. Patient differences between stimulus manipulation difficulty level and fastest response window size will provide improvement indices to characterize each subject. All adjustments will be based on running weighted averages of trial accuracy and reaction time, continually saved/updated by the E-Prime stimulus presentation software.

**Engagement/Motivation** Cognitive training gain are believed to be optimized when patients approach trials with consistent high motivation <sup>43</sup>. We have incorporated social and minor financial incentives for engagement (rapid response time consistency) and improvements in each session. It is hoped this also will partially reduce boredom. The coach also will assess participants' subjectively-rated motivation on a 10-point Likert scale.

**Remotely-Supervised EWM Training** Our EWM training delivery is designed to maximize compliance. For a typical family with late middle- or high-school age children who have many, often-conflicting priorities, visits

to the Olin NRC 4 times a week for 5 weeks will impossibly compromise study feasibility. Consistent with guidelines we have proposed for other forms of remotely-supervised interventions  $^{291, 292}$ , WM training will be done 'at home' on a study-provided Lenovo TP X1 Tablet with a cellular modem and Verizon data plan. Tablets will run GoToAssist's 'RemoteDesktop' software so Olin NRC staff can remotely administer EWM practice sessions. Study staff can remotely start the session (even when the tablet is powered down), initiate Skype videoconferencing for a 'virtual presence' during training, and load pre-configured E-Prime EWM task training exercises. Training behavioral data are transferred daily to Olin NRC servers for archiving via FTP. Each tablet is password-locked and will run Absolute software that provides GPS location and the ability to erase all data in case of loss or theft. We successfully used these procedures for our n=7 EWM training ADHD pilot study. This, and our other success with supervised ADHD WM training  $^{103}$ , validates the feasibility of the novel training delivery approach. *Coaching* During each session, a project staff member will interact with each participant through this virtual connection. As in other types of WM training, such a 'coach' works closely with families to help problem-solve unanticipated barriers to regular practice.

R61 and R33 Hypothesis-Testing General Comments Missing data bias tests will use Little's multivariate test, as well as univariate counterparts <sup>293</sup>. Missing data will be dealt with using Full Information Maximum Likelihood algorithms <sup>294</sup> or pattern mixture modeling, as appropriate <sup>295</sup>. Outlier and specification error diagnostics will be examined. All data will be examined to ensure they meet statistical test assumptions. If not, we will use robust estimators based either on Huber-White estimation, bootstrapping, or methods described in Wilcox <sup>296</sup>. Group fMRI analyses will use PALM <sup>297</sup> – a CIFTI data format-compatible analysis tool that applies threshold-free cluster enhancement for surface-based fMRI analysis and multiple comparisons corrections with permutation-based inference. All group analyses will use age as a covariate to account for any maturational differences. We will examine sex differences as per NOT-OD-15-102.

R33 Goals The 3-year R33 study will seek to replicate R61 target engagement evidence in a larger sample, using analyses robust to factors that potentially might mitigate outcomes. It also will determine if EWM training target engagement can be linked to clinically-relevant behavioral change. We do not intend the R33 to be a formal efficacy test; it is intended only to inform a decision about the potential of an EWM training intervention for a subsequent efficacy trial testing. Secondary goals are to inform the design of possible future efficacy studies by a) learning if ADHD EWM gains represent resolution of brain function deficits compared to non-ADHD, assessed by recruiting a demographically-matched n=40 non-ADHD comparison adolescent sample who will undergo 2 evaluations, also  $\sim$ 5 weeks apart, b) determining whether EWM gains generalize to non-

trained EWM tasks, c) examining the effect of intervention non-adherence on target engagement, and d) identifying ADHD characteristics that might moderate EWM training outcomes which could influence the design of subsequent efficacy research.

Gene Banking We envision a need to have whole-genome data in this richly phenotyped dataset to answer emerging questions. Saliva sampling costs were budgeted and samples will be stored at Olin for future use.

R33 Trial Methodology The R33 will use the same R61 EWM training intervention. As such, it will have the same randomization, coaching, discontinuation rules, allocation concealment, 5-week baseline/endpoint assessment timeframe, target 'dose' of 20-25 EWM training or 'sham training' placebo sessions, and www.clinicaltrials.gov registration. After 20%

Assessed for Enrollment eligibility (N=150)  $\mathbf{V}$ Randomized (n=90)Allocation EWM Active Training Placebo (n=45)(n=45)Endpoint 5 Week Completers Completers for Analysis for Analysis (n=36)(n=36)Fig 11. R33 CONSORT diagram

expected attrition, there should be 36 ADHD 'completers' in each arm (Fig. 11). Unlike the R61, the R33 also will examine a primary clinical endpoint (ADHD symptom severity) and secondary outcomes (3 psychosocial function assessment measurements; see Table 1). The R33 also will formally evaluate <u>Training Non-Adherence</u> using CACE analyses of compliance effects <sup>300</sup> on target engagement. We define 'protocol non-adherence' as <80% session completion, with the goal of at least 20 sessions by an endpoint 5 weeks after trial start. Any change to a participant's type/dose of medications or adding another form of treatment (e.g., neurofeedback, etc.) also will be non-compliance. 'Procedural non-adherence' is defined as poor quality engagement, as rated both subjectively and objectively by the training coach via virtual observation of each session (see appended Intervention Manual).

R33 Hypothesis-Testing We remind reviewers PHS-CT supplement Section 4 contains the detailed hypothesis-testing plan, including several important supplemental analyses to greatly enhance study impact.

R33 Power Analysis Power for this study's ANCOVA analyses of treatment outcome is primarily impacted by three factors -1) sample size, 2) effect size d, and 3) the strength of association  $R^2$  between the dependent variable and any model covariates. Figure 12 shows ANCOVA power analysis estimates for the expected 81 of 90 R33 completers. We see power will be at or greater than 80% for Cohen's d > 0.57 effect sizes for any ANCOVA test where the  $R^2$  for the covariate terms alone falls above 0.16. These anticipated  $R^2$  values we tested are realistic. Quantile analysis found a convincing majority (85%) of the R<sup>2</sup> distribution values across all the R61 trial's functional connectivity ANCOVA models were well above 0.16. In sum, the R33 design is adequately powered for a credible replication study. Its power will suffice to confirm R61 findings even if the new R33 ADHD sample shows the same result at a slightly lower effect size magnitude. Alternatively, we could decrease α to .01 for any specific brain connectivity replication test while maintaining sensitivity to a comparable d = 0.68 effect size magnitude



(i.e., approximately the same as the smallest effects reported in the R61).

R33 Impact on Decision to Continue Research The R33 phase results will inform a decision about whether the intervention shows potential for improving clinical outcomes. A large-scale efficacy trial will be recommended only if a) R61 behavioral and biological target engagement evidence is replicated in the new R33 ADHD sample, and b) if there is evidence for a meaningful association between EWM training-induced target engagement and credible ADHD clinical changes over the brief 5-week R33 trial. The magnitude of any clinical changes (great or small) also will be instructive in deciding whether or not this intervention development research should advance in future studies to efficacy testing. Moreover, the specific endpoints that show improvement will be the focus of any subsequent RCT proposal. Secondary R33 analyses will confirm the remotely-supervised EWM training approach has the anticipated acceptability, tolerability, and retention.

### **Key Study Design Choices to Maximize Robust Results**

- 1) Sample Sizes Careful statistical power analyses were done to support adequate sampling for confidence that both R61 and R33 phase results would provide a definitive Yes/No answers about target engagement.
- 2) <u>Use of Placebo Control</u> Both R61 and R33 include random assignment to placebo for strongest inference possible about whether target engagement is due to the intervention. Moreover, the behavioral and neural targets are objective and likely robust to any expectancy effects seen in prior research.
- 3) How To Handle ADHD WM Deficits Pre-existing cognitive ability has an equivocal relationship to training-related cognitive gains 301-303 and there is no published guidance as to what effect ADHD deficits might have on training outcomes. As such, our R33 will ensure any evidence for target engagement is robust to sample variability in pre-training EWM ability levels.
- 4) Other ADHD Clinical Heterogeneity There are many ADHD clinical characteristics (co-morbidities, medication histories, etc.) and suspected etiological biomarkers (including variable WM expression) that might influence EWM target engagement. If the R61/R33 is successful, supplemental analyses will begin to assess possible moderation effects to inform future sampling plans and research design.
- 5) <u>EWM Tasks for Training vs. Brain Target Assessment?</u> The only way to be confident neural target engagement reflects EWM training effects is to use the exact same tasks for both fMRI and training. However, it remains important to show EWM is training actual 'ability' and not just maximizing specific task performance. As such, we will examine 'near transfer' of training gains to 4 non-trained EWM *Shifting*, *Updating*, *Distractor Filtering* and *Suppression* tests (Table 2). We also will conduct exploratory 'far transfer' analyses of simple WM short-term storage and any training effects on other executive function <sup>304-306</sup> tasks.
- 6) <u>Interpretation of EWM Training Effects</u> We will compare ADHD training effects to data from non-ADHD participants to better understand trial outcomes. We are open to the possibility that brain changes either

- resolve abnormalities, or alternatively that they build upon intact neural systems to enhance ability, thereby 'compensating' for other deficits. Either underlying mechanism would support future efficacy research.
- 7) <u>Theoretical Advances</u> PHS-CT Section 4 describes several supplemental analyses using pooled R61 and R33 trial outcome data that might refine our conceptual model of how the EWM intervention works.

Other Study Design Features For Rigor/Reproducibility This R61/R33 provides a built-in replication by design. We use strong RCT design principles and we avoid many methodological pitfalls of prior ADHD WM training RCTs. We base sampling attrition estimates on direct experience to ensure our final sample size will be adequate; statistical power was carefully confirmed for our planned hypothesis-testing, using conservative estimates. Only a small handful of treatment targets will be tested for engagement, requiring a very specific, narrow path towards study milestone achievement. The R61 and R33 use the same intervention to ensure continuity between the two study phases. Protocol compliance will be closely monitored and its effects on target engagement will be formally evaluated in the R33 analysis plan. Clinical and cognitive tests have high test-retest reliability and are validated for adolescents. We use well-validated, piloted fMRI tasks with rigorous QC procedures to obtain high-quality, movement free MRI data. HCP methods offer the most accurate localization of brain function. We avoid the interpretive confounds of assessing ADHD patients' EWM ability when they are medicated. Data will be made available in NDA repositories so other investigators will be free to re-examine our results, or extend findings with new analyses.

#### References

- 1. Association, A.P., *Diagnostic and statistical manual of mental disorders*. 5th ed2013, Arlington, VA: American Psychiatric Publishing.
- 2. Biederman, J., *Attention-deficit/hyperactivity disorder: a life-span perspective*. J Clin Psychiatry, 1998. **59 Suppl 7**: p. 4-16.
- 3. Kessler, R.C., L. Adler, R. Barkley, J. Biederman, C.K. Conners, O. Demler, S.V. Faraone, L.L. Greenhill, M.J. Howes, K. Secnik, T. Spencer, T.B. Ustun, E.E. Walters, and A.M. Zaslavsky, *The prevalence and correlates of adult ADHD in the United States: results from the National Comorbidity Survey Replication*. Am J Psychiatry, 2006. **163**(4): p. 716-23.
- 4. Barkley, R.A., M. Fischer, L. Smallish, and K. Fletcher, *The persistence of attention-deficit/hyperactivity disorder into young adulthood as a function of reporting source and definition of disorder*. J Abnorm Psychol, 2002. **111**(2): p. 279-89.
- 5. Barkley, R.A., M. Fischer, L. Smallish, and K. Fletcher, *Young adult outcome of hyperactive children:* adaptive functioning in major life activities. J Am Acad Child Adolesc Psychiatry, 2006. **45**(2): p. 192-202.
- 6. Breslau, J., E. Miller, N. Breslau, K. Bohnert, V. Lucia, and J. Schweitzer, *The impact of early behavior disturbances on academic achievement in high school.* Pediatrics, 2009. **123**(6): p. 1472-6. **PMCID**: 2778327
- 7. Breslau, J., E. Miller, W.J. Joanie Chung, and J.B. Schweitzer, *Childhood and adolescent onset psychiatric disorders*, *substance use*, *and failure to graduate high school on time*. J Psychiatr Res, 2011. **45**(3): p. 295-301. **PMCID**: 2962709
- 8. Hinshaw, S.P., *Academic underachievement, attention deficits, and aggression: comorbidity and implications for intervention.* J Consult Clin Psychol, 1992. **60**(6): p. 893-903.
- 9. Hinshaw, S.P., *Externalizing behavior problems and academic underachievement in childhood and adolescence: causal relationships and underlying mechanisms.* Psychol Bull, 1992. **111**(1): p. 127-55.
- 10. Polderman, T.J., D.I. Boomsma, M. Bartels, F.C. Verhulst, and A.C. Huizink, *A systematic review of prospective studies on attention problems and academic achievement*. Acta Psychiatr Scand, 2010. **122**(4): p. 271-84.
- 11. Raggi, V.L. and A.M. Chronis, *Interventions to address the academic impairment of children and adolescents with ADHD*. Clin Child Fam Psychol Rev, 2006. **9**(2): p. 85-111.
- Wilens, T.E., Attention-deficit/hyperactivity disorder and the substance use disorders: the nature of the relationship, subtypes at risk, and treatment issues. Psychiatr Clin North Am, 2004. **27**(2): p. 283-301.
- 13. Levin, F.R., S.M. Evans, and H.D. Kleber, *Prevalence of adult attention-deficit hyperactivity disorder among cocaine abusers seeking treatment*. Drug Alcohol Depend, 1998. **52**(1): p. 15-25.
- 14. Molina, B.S., S.P. Hinshaw, J.M. Swanson, L.E. Arnold, B. Vitiello, P.S. Jensen, J.N. Epstein, B. Hoza, L. Hechtman, H.B. Abikoff, G.R. Elliott, L.L. Greenhill, J.H. Newcorn, K.C. Wells, T. Wigal, R.D. Gibbons, K. Hur, P.R. Houck, and M.T.A.C. Group, *The MTA at 8 years: prospective follow-up of children treated for combined-type ADHD in a multisite study*. J Am Acad Child Adolesc Psychiatry, 2009. **48**(5): p. 484-500. **PMCID**: 3063150
- Jensen, P.S., L.E. Arnold, J.M. Swanson, B. Vitiello, H.B. Abikoff, L.L. Greenhill, L. Hechtman, S.P. Hinshaw, W.E. Pelham, K.C. Wells, C.K. Conners, G.R. Elliott, J.N. Epstein, B. Hoza, J.S. March, B.S. Molina, J.H. Newcorn, J.B. Severe, T. Wigal, R.D. Gibbons, and K. Hur, *3-year follow-up of the NIMH MTA study*. J Am Acad Child Adolesc Psychiatry, 2007. **46**(8): p. 989-1002.
- 16. A 14-month randomized clinical trial of treatment strategies for attention-deficit/hyperactivity disorder. The MTA Cooperative Group. Multimodal Treatment Study of Children with ADHD. Arch Gen Psychiatry, 1999. **56**(12): p. 1073-86.
- 17. Pliszka, S. and A.W.G.o.Q. Issues, *Practice parameter for the assessment and treatment of children and adolescents with attention-deficit/hyperactivity disorder*. J Am Acad Child Adolesc Psychiatry, 2007. **46**(7): p. 894-921.
- 18. Advokat, C., *What exactly are the benefits of stimulants for ADHD?* J Atten Disord, 2009. **12**(6): p. 495-8.
- 19. Cunningham, C.E. and R.A. Barkley, *The role of academic failure in hyperactive behavior*. J Learn Disabil, 1978. **11**(5): p. 274-80.

- 20. Barkley, R.A. and C.E. Cunningham, *Do stimulant drugs improve the academic performance of hyperkinetic children? A review of outcome studies.* Clin Pediatr (Phila), 1978. **17**(1): p. 85-92.
- Carlson, C.L. and M.R. Bunner, *Effects of methylphenidate on the academic performance of children with attention deficit hyperactive disorder and learning disabilities*. School Psychology Review, 1993. **22**: p. 184-198.
- 22. Loe, I.M. and H.M. Feldman, *Academic and educational outcomes of children with ADHD*. Ambul Pediatr, 2007. **7**(1 Suppl): p. 82-90.
- 23. Swanson, J.M., D. Cantwell, M. Lerner, K. McBurnett, and G. Hanna, *Effects of stimulant medication on learning in children with ADHD*. J Learn Disabil, 1991. **24**(4): p. 219-30, 255.
- 24. Gadow, K.D., Effects of stimulant drugs on academic performance in hyperactive and learning disabled children. J Learn Disabil, 1983. **16**(5): p. 290-9.
- 25. Greenhill, L., D.H. Beyer, J. Finkleson, D. Shaffer, J. Biederman, C.K. Conners, C. Gillberg, M. Huss, P. Jensen, J.L. Kennedy, R. Klein, J. Rapoport, T. Sagvolden, T. Spencer, J.M. Swanson, and N. Volkow, Guidelines and algorithms for the use of methylphenidate in children with Attention-Deficit/Hyperactivity Disorder. J Atten Disord, 2002. 6 Suppl 1: p. S89-100.
- 26. McLeod, J.D., B.A. Pescosolido, D.T. Takeuchi, and T.F. White, *Public attitudes toward the use of psychiatric medications for children*. J Health Soc Behav, 2004. **45**(1): p. 53-67.
- 27. Dosreis, S., J.M. Zito, D.J. Safer, K.L. Soeken, J.W. Mitchell, Jr., and L.C. Ellwood, *Parental perceptions and satisfaction with stimulant medication for attention-deficit hyperactivity disorder*. J Dev Behav Pediatr, 2003. **24**(3): p. 155-62.
- 28. Biederman, J., A.F. Arnsten, S.V. Faraone, A.E. Doyle, T.J. Spencer, T.E. Wilens, M.D. Weiss, S.A. Safren, and L. Culpepper, *New developments in the treatment of ADHD*. J Clin Psychiatry, 2006. **67**(1): p. 148-59.
- 29. Biederman, J., T.J. Spencer, T.E. Wilens, R.H. Weisler, S.C. Read, S.J. Tulloch, and S.L.I.s. group, Long-term safety and effectiveness of mixed amphetamine salts extended release in adults with ADHD. CNS Spectr, 2005. **10**(12 Suppl 20): p. 16-25.
- 30. Faraone, S.V. and H.P. Upadhyaya, *The effect of stimulant treatment for ADHD on later substance abuse and the potential for medication misuse, abuse, and diversion.* J Clin Psychiatry, 2007. **68**(11): p. e28.
- 31. Harpur, R.A., M. Thompson, D. Daley, H. Abikoff, and E.J. Sonuga-Barke, *The attention-deficit/hyperactivity disorder medication-related attitudes of patients and their parents*. J Child Adolesc Psychopharmacol, 2008. **18**(5): p. 461-73.
- Johnston, C., P. Hommersen, and C. Seipp, *Acceptability of behavioral and pharmacological treatments for attention-deficit/hyperactivity disorder: relations to child and parent characteristics.* Behav Ther, 2008. **39**(1): p. 22-32.
- 33. McCabe, S.E., C.J. Teter, and C.J. Boyd, *Medical use, illicit use and diversion of prescription stimulant medication*. J Psychoactive Drugs, 2006. **38**(1): p. 43-56. **PMCID**: 1761861
- 34. Bright, G.M., *Abuse of medications employed for the treatment of ADHD: results from a large-scale community survey.* Medscape J Med, 2008. **10**(5): p. 111. **PMCID**: 2438483
- 35. Coletti, D.J., E. Pappadopulos, N.J. Katsiotas, A. Berest, P.S. Jensen, and V. Kafantaris, *Parent perspectives on the decision to initiate medication treatment of attention-deficit/hyperactivity disorder*. J Child Adolesc Psychopharmacol, 2012. **22**(3): p. 226-37. **PMCID**: PMC3374352
- 36. Greenhill, L.L., *Clinical effects of stimulant medication in ADHD*, in *Stimulant Drugs and ADHD: Basic and Clinical Neuroscience*, M.V. Solanto, A.F.T. Arnsten, and F.X. Castellanos, Editors. 2001,
  Oxford University Press: New York. p. 31-57.
- 37. Visser, S.N., R.H. Bitsko, M.L. Danielson, R. Gandhour, S.J. Blumberg, L. Schieve, J. Holbrook, M. Wolraich, and S. Cuffe, *Treatment of attention-deficit/hyperactivity disorder among children with special health care needs*. Journal of Pediatrics.
- 38. Prevalence of diagnosis and medication treatment for Attention-Deficit/Hyperactivity Disorder United States, 2003, D.o.H.a.H. Services., Editor 2005, Centers for Disease Control. p. 841-847.
- 39. Doshi, J.A., P. Hodgkins, J. Kahle, V. Sikirica, M.J. Cangelosi, J. Setyawan, M.H. Erder, and P.J. Neumann, *Economic impact of childhood and adult attention-deficit/hyperactivity disorder in the United States*. J Am Acad Child Adolesc Psychiatry, 2012. **51**(10): p. 990-1002 e2.
- 40. Klingberg, T., H. Forssberg, and H. Westerberg, *Training of working memory in children with ADHD*. J Clin Exp Neuropsychol, 2002. **24**(6): p. 781-91.

- 41. Pascual-Leone, A., A. Amedi, F. Fregni, and L.B. Merabet, *The plastic human brain cortex*. Annu Rev Neurosci, 2005. **28**: p. 377-401.
- 42. Guida, A., F. Gobet, and S. Nicolas, Functional cerebral reorganization: a signature of expertise? Reexamining Guida, Gobet, Tardieu, and Nicolas' (2012) two-stage framework. Front Hum Neurosci, 2013. 7: p. 590. **PMCID**: 3778237
- 43. Vinogradov, S., M. Fisher, and E. de Villers-Sidani, *Cognitive training for impaired neural systems in neuropsychiatric illness.* Neuropsychopharmacology, 2012. **37**(1): p. 43-76. **PMCID**: PMC3238091
- 44. Caeyenberghs, K., A. Clemente, P. Imms, G. Egan, D.R. Hocking, A. Leemans, C. Metzler-Baddeley, D.K. Jones, and P.H. Wilson, *Evidence for Training-Dependent Structural Neuroplasticity in Brain-Injured Patients: A Critical Review*. Neurorehabil Neural Repair, 2018. **32**(2): p. 99-114.
- 45. Hamaide, J., G. De Groof, and A. Van der Linden, *Neuroplasticity and MRI: A perfect match*. Neuroimage, 2016. **131**: p. 13-28.
- 46. Merzenich, M.M., T.M. Van Vleet, and M. Nahum, *Brain plasticity-based therapeutics*. Front Hum Neurosci, 2014. **8**: p. 385. **PMCID**: PMC4072971
- 47. Nahum, M., H. Lee, and M.M. Merzenich, *Principles of neuroplasticity-based rehabilitation*. Prog Brain Res, 2013. **207**: p. 141-71.
- 48. Nguyen, L., K. Murphy, and G. Andrews, *Cognitive and neural plasticity in old age: A systematic review of evidence from executive functions cognitive training*. Ageing Res Rev, 2019. **53**: p. 100912.
- 49. Park, D.C. and G.N. Bischof, *The aging mind: neuroplasticity in response to cognitive training*. Dialogues Clin Neurosci, 2013. **15**(1): p. 109-19. **PMCID**: PMC3622463
- 50. Qi, X.L. and C. Constantinidis, *Neural changes after training to perform cognitive tasks*. Behav Brain Res, 2013. **241**: p. 235-43. **PMCID**: PMC3552071
- 51. Walhovd, K.B., R. Westerhausen, A.M. de Lange, A.C. Brathen, H. Grydeland, A. Engvig, and A.M. Fjell, *Premises of plasticity And the loneliness of the medial temporal lobe*. Neuroimage, 2016. **131**: p. 48-54.
- 52. Chein, J.M. and A.B. Morrison, *Expanding the mind's workspace: training and transfer effects with a complex working memory span task.* Psychon Bull Rev, 2010. **17**(2): p. 193-9.
- 53. Klingberg, T., E. Fernell, P.J. Olesen, M. Johnson, P. Gustafsson, K. Dahlstrom, C.G. Gillberg, H. Forssberg, and H. Westerberg, *Computerized training of working memory in children with ADHD--a randomized, controlled trial.* J Am Acad Child Adolesc Psychiatry, 2005. **44**(2): p. 177-86.
- 54. Cowan, N., E.M. Elliott, J. Scott Saults, C.C. Morey, S. Mattox, A. Hismjatullina, and A.R. Conway, *On the capacity of attention: its estimation and its role in working memory and cognitive aptitudes.* Cogn Psychol, 2005. **51**(1): p. 42-100. **PMCID**: 2673732
- 55. Engle, R.W., S.W. Tuholski, J.E. Laughlin, and A.R. Conway, *Working memory, short-term memory, and general fluid intelligence: a latent-variable approach.* J Exp Psychol Gen, 1999. **128**(3): p. 309-31.
- Oberauer, K., R. Schulze, O. Wilhelm, and H.M. Suss, *Working memory and intelligence--their correlation and their relation: comment on Ackerman, Beier, and Boyle (2005).* Psychol Bull, 2005. **131**(1): p. 61-5; author reply 72-5.
- 57. Kane, M.J., D.Z. Hambrick, S.W. Tuholski, O. Wilhelm, T.W. Payne, and R.W. Engle, *The generality of working memory capacity: a latent-variable approach to verbal and visuospatial memory span and reasoning*. J Exp Psychol Gen, 2004. **133**(2): p. 189-217.
- 58. Turner, M.L. and R.W. Engle, *Is woring memory capcity task dependent?* Journal of Memory and Language, 1989. **28**(127-154).
- 59. Daneman, M. and P.A. Carpenter, *Individual differences in working memory and reading*. Journal of Verbal learning & Verbal Behaviora, 1980. **19**(450-466).
- 60. Gathercole, S.E. and S.J. Pickering, *Working memory deficits in children with low achievements in the national curriculum at 7 years of age*. Br J Educ Psychol, 2000. **70 (Pt 2)**: p. 177-94.
- 61. Swanson, H.L. and M. Beebe-Frankenberger, *The relationship between working memory and mathematical problem solving in children at risk and not at risk for math disabilities*. Journal of Education Psychology, 2004. **96**(471-491).
- 62. Swanson, H.L. and O. Jerman, *The influence of working memory on reading growth in subgroups of children with reading disabilities*. J Exp Child Psychol, 2007. **96**(4): p. 249-83.
- 63. Swanson, H.L., O. Jerman, and X. Zheng, *Growth in working memory and mathematic problem solving in children at risk and not at risk for serious math difficulties*. Journal of Educational Psychology, 2008. **100**(343-379).

- 64. Fried, R., J. Chan, L. Feinberg, A. Pope, K.Y. Woodworth, S.V. Faraone, and J. Biederman, *Clinical correlates of working memory deficits in youth with and without ADHD: A controlled study.* J Clin Exp Neuropsychol, 2016. **38**(5): p. 487-96. **PMCID**: PMC4970465
- 65. Kofler, M.J., D.E. Sarver, J.A. Spiegel, T.N. Day, S.L. Harmon, and E.L. Wells, *Heterogeneity in ADHD:* Neurocognitive predictors of peer, family, and academic functioning. Child Neuropsychol, 2016: p. 1-27.
- ota van Lieshout, M., M. Luman, J.W. Twisk, S.V. Faraone, D.J. Heslenfeld, C.A. Hartman, P.J. Hoekstra, B. Franke, J.K. Buitelaar, N.N. Rommelse, and J. Oosterlaan, *Neurocognitive Predictors of ADHD Outcome: a 6-Year Follow-up Study.* J Abnorm Child Psychol, 2016.
- 67. Buhner, M., C.J. König, M. Prick, and S. Krumm, *Working memory dimensions as differential predictors of the speed and error aspect of multitasking performance*. Human Performance, 2006. **19**(253-275).
- 68. Hambrick, D.Z., F.L. Oswald, E.S. Darowski, T.A. Rench, and R. Brou, *Predictors of multitasking performance in a synthetic work paradigm*. Applied Cognitive Psychology, 2010. **24**(1149-1167).
- 69. Kane, M.J., L.H. Brown, J.C. McVay, P.J. Silvia, I. Myin-Germeys, and T.R. Kwapil, For whom the mind wanders, and when: an experience-sampling study of working memory and executive control in daily life. Psychol Sci, 2007. **18**(7): p. 614-21.
- 70. Engle, R.W., J.J. Carullo, and K.W. Collins, *Individual differences in the role of working memory in comprehension and following directions*. Journal of Educational Research, 1991. **84**(253-262).
- 71. Gathercole, S.E., E. Durling, M. Evans, S. Jeffcock, and S. Stone, *Working memory deficits in laboratory analogues of activities*. Applied Cognitive Psychology, 2008. **22**(1019-1037).
- 72. Kasper, L.J., R.M. Alderson, and K.L. Hudec, *Moderators of working memory deficits in children with attention-deficit/hyperactivity disorder (ADHD): a meta-analytic review.* Clin Psychol Rev, 2012. **32**(7): p. 605-17.
- 73. Martinussen, R., J. Hayden, S. Hogg-Johnson, and R. Tannock, *A meta-analysis of working memory impairments in children with attention-deficit/hyperactivity disorder*. J Am Acad Child Adolesc Psychiatry, 2005. **44**(4): p. 377-84.
- 74. Doyle, A.E., *Executive functions in attention-deficit/hyperactivity disorder*. J Clin Psychiatry, 2006. **67 Suppl 8**: p. 21-6.
- 75. Ramos, A.A., A.C. Hamdan, and L. Machado, *A meta-analysis on verbal working memory in children and adolescents with ADHD.* Clin Neuropsychol, 2019: p. 1-26.
- 76. Rubia, K., Cognitive Neuroscience of Attention Deficit Hyperactivity Disorder (ADHD) and Its Clinical Translation. Front Hum Neurosci, 2018. **12**: p. 100. **PMCID**: 5884954
- 77. Willcutt, E.G., A.E. Doyle, J.T. Nigg, S.V. Faraone, and B.F. Pennington, *Validity of the executive function theory of attention-deficit/hyperactivity disorder: a meta-analytic review.* Biol Psychiatry, 2005. **57**(11): p. 1336-46.
- 78. Alderson, R.M., L.J. Kasper, K.L. Hudec, and C.H. Patros, *Attention-deficit/hyperactivity disorder* (*ADHD*) and working memory in adults: a meta-analytic review. Neuropsychology, 2013. **27**(3): p. 287-302.
- 79. Arnsten, A.F., Toward a new understanding of attention-deficit hyperactivity disorder pathophysiology: an important role for prefrontal cortex dysfunction. CNS Drugs, 2009. **23 Suppl 1**: p. 33-41.
- 80. Pievsky, M.A. and R.E. McGrath, *Neurocognitive effects of methylphenidate in adults with attention-deficit/hyperactivity disorder: A meta-analysis.* Neurosci Biobehav Rev, 2018. **90**: p. 447-455.
- 81. Pievsky, M.A. and R.E. McGrath, *The Neurocognitive Profile of Attention-Deficit/Hyperactivity Disorder: A Review of Meta-Analyses*. Arch Clin Neuropsychol, 2018. **33**(2): p. 143-157.
- 82. Schwarz, E., H. Tost, and A. Meyer-Lindenberg, *Working memory genetics in schizophrenia and related disorders: An RDoC perspective*. Am J Med Genet B Neuropsychiatr Genet, 2016. **171B**(1): p. 121-31.
- 83. Sonuga-Barke, E.J., S. Cortese, G. Fairchild, and A. Stringaris, *Annual Research Review:*Transdiagnostic neuroscience of child and adolescent mental disorders--differentiating decision making in attention-deficit/hyperactivity disorder, conduct disorder, depression, and anxiety. J Child Psychol Psychiatry, 2016. **57**(3): p. 321-49. **PMCID**: PMC4762324

- 84. van Amelsvoort, T. and D. Hernaus, Effect of Pharmacological Interventions on the Fronto-Cingulo-Parietal Cognitive Control Network in Psychiatric Disorders: A Transdiagnostic Systematic Review of fMRI Studies. Front Psychiatry, 2016. 7: p. 82. PMCID: PMC4870274
- 85. Nigg, J.T., H.C. Gustafsson, S.L. Karalunas, P. Ryabinin, S.K. McWeeney, S.V. Faraone, M.A. Mooney, D.A. Fair, and B. Wilmot, *Working Memory and Vigilance as Multivariate Endophenotypes Related to Common Genetic Risk for Attention-Deficit/Hyperactivity Disorder*. J Am Acad Child Adolesc Psychiatry, 2018. **57**(3): p. 175-182. **PMCID**: PMC6547382
- 86. Vuijk, P.J., J. Martin, E.B. Braaten, G. Genovese, M.R. Capawana, S.M. O'Keefe, B.A. Lee, H.S. Lind, J.W. Smoller, S.V. Faraone, R.H. Perlis, and A.E. Doyle, *Translating Discoveries in Attention-Deficit/Hyperactivity Disorder Genomics to an Outpatient Child and Adolescent Psychiatric Cohort.* J Am Acad Child Adolesc Psychiatry, 2019.
- 87. Sudre, G., J. Frederick, W. Sharp, A. Ishii-Takahashi, A. Mangalmurti, S. Choudhury, and P. Shaw, Mapping associations between polygenic risks for childhood neuropsychiatric disorders, symptoms of attention deficit hyperactivity disorder, cognition, and the brain. Mol Psychiatry, 2019. **PMCID**: PMC6667324
- 88. Martin, J., M.L. Hamshere, E. Stergiakouli, M.C. O'Donovan, and A. Thapar, *Neurocognitive abilities in the general population and composite genetic risk scores for attention-deficit hyperactivity disorder*. J Child Psychol Psychiatry, 2015. **56**(6): p. 648-56. **PMCID**: PMC4431584
- 89. Buschkuehl, M., S.M. Jaeggi, and J. Jonides, *Neuronal effects following working memory training*. Dev Cogn Neurosci, 2012. **2 Suppl 1**: p. S167-79.
- 90. Brehmer, Y., H. Westerberg, and L. Backman, *Working-memory training in younger and older adults:* training gains, transfer, and maintenance. Front Hum Neurosci, 2012. **6**: p. 63. **PMCID**: 3313479
- Jolles, D.D., M.J. Grol, M.A. Van Buchem, S.A. Rombouts, and E.A. Crone, *Practice effects in the brain: Changes in cerebral activation after working memory practice depend on task demands.* Neuroimage, 2010. **52**(2): p. 658-68.
- 92. Hempel, A., F.L. Giesel, N.M. Garcia Caraballo, M. Amann, H. Meyer, T. Wustenberg, M. Essig, and J. Schroder, *Plasticity of cortical activation related to working memory during training*. Am J Psychiatry, 2004. **161**(4): p. 745-7.
- 93. Olesen, P.J., H. Westerberg, and T. Klingberg, *Increased prefrontal and parietal activity after training of working memory*. Nat Neurosci, 2004. **7**(1): p. 75-9.
- 94. Westerberg, H. and T. Klingberg, *Changes in cortical activity after training of working memory--a single-subject analysis*. Physiol Behav, 2007. **92**(1-2): p. 186-92.
- 95. Heinzel, S., R.C. Lorenz, W.R. Brockhaus, T. Wustenberg, N. Kathmann, A. Heinz, and M.A. Rapp, Working memory load-dependent brain response predicts behavioral training gains in older adults. J Neurosci, 2014. **34**(4): p. 1224-33.
- 96. Strenziok, M., R. Parasuraman, E. Clarke, D.S. Cisler, J.C. Thompson, and P.M. Greenwood, *Neurocognitive enhancement in older adults: comparison of three cognitive training tasks to test a hypothesis of training transfer in brain connectivity.* Neuroimage, 2014. **85 Pt 3**: p. 1027-39.
- 97. Takeuchi, H., Y. Taki, R. Nouchi, H. Hashizume, A. Sekiguchi, Y. Kotozaki, S. Nakagawa, C.M. Miyauchi, Y. Sassa, and R. Kawashima, *Effects of working memory training on functional connectivity and cerebral blood flow during rest*. Cortex, 2013. **49**(8): p. 2106-25.
- 98. Langer, N., C.C. von Bastian, H. Wirz, K. Oberauer, and L. Jancke, *The effects of working memory training on functional brain network efficiency*. Cortex, 2013. **49**(9): p. 2424-38.
- 99. Broyd, S.J., C. Demanuele, S. Debener, S.K. Helps, C.J. James, and E.J. Sonuga-Barke, *Default-mode brain dysfunction in mental disorders: a systematic review*. Neuroscience & Biobehavioral Reviews, 2009. **33**(3): p. 279-96.
- 100. Anticevic, A., M.W. Cole, J.D. Murray, P.R. Corlett, X.J. Wang, and J.H. Krystal, *The role of default network deactivation in cognition and disease*. Trends Cogn Sci, 2012. **16**(12): p. 584-92. **PMCID**: 3501603
- 101. Raichle, M.E. and A.Z. Snyder, *A default mode of brain function: a brief history of an evolving idea*. Neuroimage, 2007. **37**(4): p. 1083-90; discussion 1097-9.
- 102. Whitfield-Gabrieli, S. and J.M. Ford, *Default mode network activity and connectivity in psychopathology*. Annu Rev Clin Psychol, 2012. **8**: p. 49-76.

- 103. Stevens, M.C., A. Gaynor, K.L. Bessette, and G.D. Pearlson, *A preliminary study of the effects of working memory training on brain function*. Brain Imaging Behav, 2016. **10**(2): p. 387-407. **PMCID**: PMC4698365
- 104. Prehn-Kristensen, A., K. Krauel, H. Hinrichs, J. Fischer, U. Malecki, H. Schuetze, S. Wolff, O. Jansen, E. Duezel, and L. Baving, *Methylphenidate does not improve interference control during a working memory task in young patients with attention-deficit hyperactivity disorder*. Brain Res, 2011. **1388**: p. 56-68.
- 105. Vance, A., T.J. Silk, M. Casey, N.J. Rinehart, J.L. Bradshaw, M.A. Bellgrove, and R. Cunnington, *Right* parietal dysfunction in children with attention deficit hyperactivity disorder, combined type: a functional MRI study. Mol Psychiatry, 2007. **12**(9): p. 826-32, 793.
- 106. Wolf, R.C., M.M. Plichta, F. Sambataro, A.J. Fallgatter, C. Jacob, K.P. Lesch, M.J. Herrmann, C. Schonfeldt-Lecuona, B.J. Connemann, G. Gron, and N. Vasic, *Regional brain activation changes and abnormal functional connectivity of the ventrolateral prefrontal cortex during working memory processing in adults with attention-deficit/hyperactivity disorder*. Hum Brain Mapp, 2009. **30**(7): p. 2252-66.
- 107. Chacko, A., N. Feirsen, A.C. Bedard, D. Marks, J.Z. Uderman, and A. Chimiklis, *Cogmed Working Memory Training for youth with ADHD: a closer examination of efficacy utilizing evidence-based criteria*. J Clin Child Adolesc Psychol, 2013. **42**(6): p. 769-83. **PMCID**: 3744604
- 108. Evans, S.W., J.S. Owens, and N. Bunford, *Evidence-Based Psychosocial Treatments for Children and Adolescents with Attention-Deficit/Hyperactivity Disorder*. J Clin Child Adolesc Psychol, 2013.
- 109. Morrison, A.B. and J.M. Chein, *Does working memory training work? The promise and challenges of enhancing cognition by training working memory.* Psychon Bull Rev, 2011. **18**(1): p. 46-60.
- Rutledge, K.J., W. van den Bos, S.M. McClure, and J.B. Schweitzer, *Training cognition in ADHD:* current findings, borrowed concepts, and future directions. Neurotherapeutics, 2012. **9**(3): p. 542-58. **PMCID**: 3441933
- 111. Shipstead, Z., K.L. Hicks, and R.W. Engle, *Cogmed working memory training: Does the evidence support the claims?* Journal of Applied Research in Memory and Cognition, 2012. **1**: p. 185-193.
- Shipstead, Z., T.S. Redick, and R.W. Engle, *Is working memory training effective?* Psychol Bull, 2012. **138**(4): p. 628-54.
- Toplak, M.E., L. Connors, J. Shuster, B. Knezevic, and S. Parks, *Review of cognitive, cognitive-behavioral, and neural-based interventions for Attention-Deficit/Hyperactivity Disorder (ADHD)*. Clin Psychol Rev, 2008. **28**(5): p. 801-23.
- 114. Hodgson, K., A.D. Hutchinson, and L. Denson, *Nonpharmacological Treatments for ADHD: A Meta-Analytic Review*. J Atten Disord, 2012.
- 115. Melby-Lervag, M. and C. Hulme, *Is working memory training effective? A meta-analytic review*. Dev Psychol, 2013. **49**(2): p. 270-91.
- 116. Rapport, M.D., S.A. Orban, M.J. Kofler, and L.M. Friedman, *Do programs designed to train working memory, other executive functions, and attention benefit children with ADHD? A meta-analytic review of cognitive, academic, and behavioral outcomes.* Clin Psychol Rev, 2013. **33**(8): p. 1237-52.
- 117. Sonuga-Barke, E.J., D. Brandeis, S. Cortese, D. Daley, M. Ferrin, M. Holtmann, J. Stevenson, M. Danckaerts, S. van der Oord, M. Dopfner, R.W. Dittmann, E. Simonoff, A. Zuddas, T. Banaschewski, J. Buitelaar, D. Coghill, C. Hollis, E. Konofal, M. Lecendreux, I.C. Wong, J. Sergeant, and A.G.G. European, Nonpharmacological interventions for ADHD: systematic review and meta-analyses of randomized controlled trials of dietary and psychological treatments. Am J Psychiatry, 2013. 170(3): p. 275-89.
- Gropper, R.J., H. Gotlieb, R. Kronitz, and R. Tannock, *Working Memory Training in College Students With ADHD or LD*. J Atten Disord, 2014.
- Holmes, J., S.E. Gathercole, and D.L. Dunning, *Poor working memory: impact and interventions*. Adv Child Dev Behav, 2010. **39**: p. 1-43.
- Hovik, K.T., B.K. Saunes, A.K. Aarlien, and J. Egeland, *RCT of working memory training in ADHD:* long-term near-transfer effects. PLoS One, 2013. **8**(12): p. e80561. **PMCID**: 3857172
- Mezzacappa, E. and J.C. Buckner, *Working memory training for chilidren with attention problems or hyperactivity: A school-based pilot study.* School Mental Health, 2010. **2**: p. 202-208.

- Gibson, B.S., D.M. Gondoli, A.C. Johnson, C.M. Steeger, B.A. Dobrzenski, and R.A. Morrissey, *Component analysis of verbal versus spatial working memory training in adolescents with ADHD: a randomized, controlled trial.* Child Neuropsychol, 2011. **17**(6): p. 546-63.
- Beck, S.J., C.A. Hanson, S.S. Puffenberger, K.L. Benninger, and W.B. Benninger, *A controlled trial of working memory training for children and adolescents with ADHD*. J Clin Child Adolesc Psychol, 2010. **39**(6): p. 825-36.
- 124. Gropper, R.J., H. Gotlieb, R. Kronitz, and R. Tannock, *Working memory training in college students with ADHD or LD*. J Atten Disord, 2014. **18**(4): p. 331-45.
- 125. Bigorra, A., M. Garolera, S. Guijarro, and A. Hervas, *Long-term far-transfer effects of working memory training in children with ADHD: a randomized controlled trial.* Eur Child Adolesc Psychiatry, 2016. **25**(8): p. 853-67.
- 126. Green, C.T., D.L. Long, D. Green, A.M. Iosif, J.F. Dixon, M.R. Miller, C. Fassbender, and J.B. Schweitzer, *Will working memory training generalize to improve off-task behavior in children with attention-deficit/hyperactivity disorder?* Neurotherapeutics, 2012. **9**(3): p. 639-48. **PMCID**: 3441930
- 127. Cortese, S., M. Ferrin, D. Brandeis, J. Buitelaar, D. Daley, R.W. Dittmann, M. Holtmann, P. Santosh, J. Stevenson, A. Stringaris, A. Zuddas, E.J. Sonuga-Barke, and A.G.G. European, *Cognitive training for attention-deficit/hyperactivity disorder: meta-analysis of clinical and neuropsychological outcomes from randomized controlled trials.* J Am Acad Child Adolesc Psychiatry, 2015. **54**(3): p. 164-74. **PMCID**: 4382075
- van Dongen-Boomsma, M., M.A. Vollebregt, D. Slaats-Willemse, and J.K. Buitelaar, [Efficacy of frequency-neurofeedback and Cogmed JM-working memory training in children with ADHD]. Tijdschr Psychiatr, 2015. **57**(7): p. 508-16.
- 129. Shuai, L., D. Daley, Y.F. Wang, J.S. Zhang, Y.T. Kong, X. Tan, and N. Ji, *Executive Function Training for Children with Attention Deficit Hyperactivity Disorder*. Chin Med J (Engl), 2017. **130**(5): p. 549-558. **PMCID**: PMC5339928
- 130. Stern, A., E. Malik, Y. Pollak, O. Bonne, and A. Maeir, *The Efficacy of Computerized Cognitive Training in Adults With ADHD: A Randomized Controlled Trial.* J Atten Disord, 2016. **20**(12): p. 991-1003.
- 131. Bikic, A., J.F. Leckman, T.O. Christensen, N. Bilenberg, and S. Dalsgaard, *Attention and executive functions computer training for attention-deficit/hyperactivity disorder (ADHD): results from a randomized, controlled trial.* Eur Child Adolesc Psychiatry, 2018. **27**(12): p. 1563-1574.
- 132. Minder, F., A. Zuberer, D. Brandeis, and R. Drechsler, *Specific Effects of Individualized Cognitive Training in Children with Attention-Deficit/Hyperactivity Disorder (ADHD): The Role of Pre-Training Cognitive Impairment and Individual Training Performance*. Dev Neurorehabil, 2019. **22**(6): p. 400-414.
- 133. Klingberg, T., *Training and plasticity of working memory*. Trends Cogn Sci, 2010. **14**(7): p. 317-24.
- Gathercole, S.E., D.L. Dunning, and J. Holmes, *Cogmed training: Let's be realistic about intervention research*. Journal of Applied Research in Memory and Cognition, 2012. **1**(3): p. 201-203.
- Rabipour, S. and A. Raz, *Training the brain: fact and fad in cognitive and behavioral remediation*. Brain Cogn, 2012. **79**(2): p. 159-79.
- 136. Takeuchi, H., Y. Taki, and R. Kawashima, *Effects of working memory training on cognitive functions and neural systems*. Rev Neurosci, 2010. **21**(6): p. 427-49.
- 137. Shah, P.J., M. Buschkuehl, S. Jaeggi, and J. Jonides, *Cognitive training for ADHD: The importance of individual differences*. Journal of Applied Research in Memory and Cognition, 2012. 1: p. 204-205.
- 138. Redick, T.S., Z. Shipstead, T.L. Harrison, K.L. Hicks, D.E. Fried, D.Z. Hambrick, M.J. Kane, and R.W. Engle, *No evidence of intelligence improvement after working memory training: a randomized, placebo-controlled study.* J Exp Psychol Gen, 2013. **142**(2): p. 359-79.
- 139. Bledowski, C., J. Kaiser, and B. Rahm, *Basic operations in working memory: contributions from functional imaging studies*. Behav Brain Res, 2010. **214**(2): p. 172-9.
- 140. Nee, D.E., J.W. Brown, M.K. Askren, M.G. Berman, E. Demiralp, A. Krawitz, and J. Jonides, *A meta-analysis of executive components of working memory*. Cereb Cortex, 2013. **23**(2): p. 264-82. **PMCID**: 3584956
- 141. Oberauer, K., *The focus of attention in working memory-from metaphors to mechanisms*. Front Hum Neurosci, 2013. **7**: p. 673. **PMCID**: PMC3797978
- 142. Harrison, T.L., Z. Shipstead, and R.W. Engle, *Why is working memory capacity related to matrix reasoning tasks?* Mem Cognit, 2015. **43**(3): p. 389-96.

- 143. Shipstead, Z., T.S. Redick, K.L. Hicks, and R.W. Engle, *The scope and control of attention as separate aspects of working memory*. Memory, 2012. **20**(6): p. 608-28.
- Engle, R.W., *Working Memory and Executive Attention: A Revisit.* Perspect Psychol Sci, 2018. **13**(2): p. 190-193.
- 145. Stoet, G., *PsyToolkit:* a software package for programming psychological experiments using Linux. Behav Res Methods, 2010. **42**(4): p. 1096-104.
- 146. Stoet, G., *PsyToolkit: A novel web-based method for running online questionnaires and reaction-time experiments.* Teaching of Psychology, 2017. **44**(1): p. 24-31.
- 147. Arechar, A.A., S. Gachter, and L. Molleman, *Conducting interactive experiments online*. Exp Econ, 2018. **21**(1): p. 99-131. **PMCID**: PMC5807491
- 148. Cunningham, J.A., A. Godinho, and V. Kushnir, *Using Mechanical Turk to recruit participants for internet intervention research: experience from recruitment for four trials targeting hazardous alcohol consumption*. BMC Med Res Methodol, 2017. **17**(1): p. 156. **PMCID**: PMC5709932
- 149. Walters, K., D.A. Christakis, and D.R. Wright, *Are Mechanical Turk worker samples representative of health status and health behaviors in the U.S.?* PLoS One, 2018. **13**(6): p. e0198835. **PMCID**: PMC5991724
- 150. Rottschy, C., R. Langner, I. Dogan, K. Reetz, A.R. Laird, J.B. Schulz, P.T. Fox, and S.B. Eickhoff, *Modelling neural correlates of working memory: a coordinate-based meta-analysis*. Neuroimage, 2012. **60**(1): p. 830-46. **PMCID**: 3288533
- 151. Anderson, M.C., K.N. Ochsner, B. Kuhl, J. Cooper, E. Robertson, S.W. Gabrieli, G.H. Glover, and J.D. Gabrieli, *Neural systems underlying the suppression of unwanted memories*. Science, 2004. **303**(5655): p. 232-5.
- Bledowski, C., B. Rahm, and J.B. Rowe, *What "works" in working memory? Separate systems for selection and updating of critical information*. J Neurosci, 2009. **29**(43): p. 13735-41. **PMCID**: PMC2785708
- 153. Butler, A.J. and K.H. James, *The neural correlates of attempting to suppress negative versus neutral memories*. Cogn Affect Behav Neurosci, 2010. **10**(2): p. 182-94.
- 154. Clapp, W.C., M.T. Rubens, and A. Gazzaley, *Mechanisms of working memory disruption by external interference*. Cereb Cortex, 2010. **20**(4): p. 859-72. **PMCID**: PMC2837090
- 155. Gazzaley, A., J. Rissman, J. Cooney, A. Rutman, T. Seibert, W. Clapp, and M. D'Esposito, *Functional interactions between prefrontal and visual association cortex contribute to top-down modulation of visual processing*. Cereb Cortex, 2007. **17 Suppl 1**: p. i125-35. **PMCID**: PMC4530799
- Johnson, M.K., C.L. Raye, K.J. Mitchell, E.J. Greene, and A.W. Anderson, *FMRI evidence for an organization of prefrontal cortex by both type of process and type of information*. Cereb Cortex, 2003. **13**(3): p. 265-73.
- Lepsien, J. and A.C. Nobre, *Attentional modulation of object representations in working memory*. Cereb Cortex, 2007. **17**(9): p. 2072-83.
- 158. Leung, H.C. and J.X. Zhang, *Interference resolution in spatial working memory*. Neuroimage, 2004. **23**(3): p. 1013-9.
- 159. McNab, F., G. Leroux, F. Strand, L. Thorell, S. Bergman, and T. Klingberg, *Common and unique components of inhibition and working memory: an fMRI, within-subjects investigation*. Neuropsychologia, 2008. **46**(11): p. 2668-82.
- 160. Mecklinger, A., K. Weber, T.C. Gunter, and R.W. Engle, *Dissociable brain mechanisms for inhibitory control: effects of interference content and working memory capacity*. Brain Res Cogn Brain Res, 2003. **18**(1): p. 26-38.
- 161. Nee, D.E. and J. Jonides, *Neural correlates of access to short-term memory*. Proc Natl Acad Sci U S A, 2008. **105**(37): p. 14228-33. **PMCID**: PMC2544606
- Nee, D.E. and J. Jonides, *Common and distinct neural correlates of perceptual and memorial selection*. Neuroimage, 2009. **45**(3): p. 963-75. **PMCID**: PMC2775536
- Nee, D.E., J. Jonides, and M.G. Berman, *Neural mechanisms of proactive interference-resolution*. Neuroimage, 2007. **38**(4): p. 740-51. **PMCID**: PMC2206737
- Nobre, A.C., J.T. Coull, P. Maquet, C.D. Frith, R. Vandenberghe, and M.M. Mesulam, *Orienting attention to locations in perceptual versus mental representations*. J Cogn Neurosci, 2004. **16**(3): p. 363-73.

- Raye, C.L., M.K. Johnson, K.J. Mitchell, J.A. Reeder, and E.J. Greene, *Neuroimaging a single thought:* dorsolateral PFC activity associated with refreshing just-activated information. Neuroimage, 2002. **15**(2): p. 447-53.
- Raye, C.L., K.J. Mitchell, J.A. Reeder, E.J. Greene, and M.K. Johnson, *Refreshing one of several active representations: behavioral and functional magnetic resonance imaging differences between young and older adults.* J Cogn Neurosci, 2008. **20**(5): p. 852-62.
- 167. Roth, J.K., M.K. Johnson, C.L. Raye, and R.T. Constable, *Similar and dissociable mechanisms for attention to internal versus external information*. Neuroimage, 2009. **48**(3): p. 601-8. **PMCID**: PMC2749565
- 168. Roth, J.K., J.T. Serences, and S.M. Courtney, *Neural system for controlling the contents of object working memory in humans*. Cereb Cortex, 2006. **16**(11): p. 1595-603.
- 169. Sorqvist, P. and B. Saetrevik, *The neural basis of updating: Distinguishing substitution processes from other concurrent processes.* Scand J Psychol, 2010. **51**(5): p. 357-62.
- 170. Toepper, M., H. Gebhardt, T. Beblo, C. Thomas, M. Driessen, M. Bischoff, C.R. Blecker, D. Vaitl, and G. Sammer, *Functional correlates of distractor suppression during spatial working memory encoding*. Neuroscience, 2010. **165**(4): p. 1244-53.
- 171. Yi, D.J., N.B. Turk-Browne, M.M. Chun, and M.K. Johnson, *When a thought equals a look: refreshing enhances perceptual memory*. J Cogn Neurosci, 2008. **20**(8): p. 1371-80. **PMCID**: PMC3213859
- 172. Zanto, T.P., M.T. Rubens, J. Bollinger, and A. Gazzaley, *Top-down modulation of visual feature* processing: the role of the inferior frontal junction. Neuroimage, 2010. **53**(2): p. 736-45. **PMCID**: PMC2930130
- 173. Zanto, T.P., M.T. Rubens, A. Thangavel, and A. Gazzaley, Causal role of the prefrontal cortex in top-down modulation of visual processing and working memory. Nat Neurosci, 2011. 14(5): p. 656-61. PMC1D: PMC3083493
- 274. Zhang, J.X., C.M. Feng, P.T. Fox, J.H. Gao, and L.H. Tan, *Is left inferior frontal gyrus a general mechanism for selection?* Neuroimage, 2004. **23**(2): p. 596-603.
- 175. Unsworth, N. and R.W. Engle, On the division of short-term and working memory: an examination of simple and complex span and their relation to higher order abilities. Psychol Bull, 2007. **133**(6): p. 1038-66.
- 176. Unsworth, N. and R.W. Engle, *The nature of individual differences in working memory capacity:* active maintenance in primary memory and controlled search from secondary memory. Psychol Rev, 2007. **114**(1): p. 104-32.
- 177. Unsworth, N. and G.J. Spillers, *Variation in working memory capacity and episodic recall: the contributions of strategic encoding and contextual retrieval.* Psychon Bull Rev, 2010. **17**(2): p. 200-5.
- 178. D'Esposito, M. and B.R. Postle, *The cognitive neuroscience of working memory*. Annu Rev Psychol, 2015. **66**: p. 115-42. **PMCID**: PMC4374359
- Heidbreder, C.A. and H.J. Groenewegen, *The medial prefrontal cortex in the rat: evidence for a dorso-ventral distinction based upon functional and anatomical characteristics*. Neurosci Biobehav Rev, 2003. **27**(6): p. 555-79.
- 180. Rosenkilde, C.E., Functional heterogeneity of the prefrontal cortex in the monkey: a review. Behav Neural Biol, 1979. **25**(3): p. 301-45.
- 181. Levy, B.J. and A.D. Wagner, *Cognitive control and right ventrolateral prefrontal cortex: reflexive reorienting, motor inhibition, and action updating.* Ann N Y Acad Sci, 2011. **1224**: p. 40-62. **PMCID**: PMC3079823
- 182. Zald, D.H. and C. Andreotti, *Neuropsychological assessment of the orbital and ventromedial prefrontal cortex*. Neuropsychologia, 2010. **48**(12): p. 3377-91.
- 183. D'Esposito, M., B.R. Postle, and B. Rypma, *Prefrontal cortical contributions to working memory:* evidence from event-related fMRI studies. Exp Brain Res, 2000. **133**(1): p. 3-11.
- 184. Petrides, M., Dissociable roles of mid-dorsolateral prefrontal and anterior inferotemporal cortex in visual working memory. J Neurosci, 2000. **20**(19): p. 7496-503.
- 185. Smith, E.E. and J. Jonides, *Storage and executive processes in the frontal lobes*. Science, 1999. **283**(5408): p. 1657-61.
- 186. Funahashi, S., C.J. Bruce, and P.S. Goldman-Rakic, *Mnemonic coding of visual space in the monkey's dorsolateral prefrontal cortex*. J Neurophysiol, 1989. **61**(2): p. 331-49.

- 187. Fuster, J.M. and G.E. Alexander, *Neuron activity related to short-term memory*. Science, 1971. **173**(3997): p. 652-4.
- 188. Miller, E.K., C.A. Erickson, and R. Desimone, *Neural mechanisms of visual working memory in prefrontal cortex of the macaque*. J Neurosci, 1996. **16**(16): p. 5154-67.
- 189. Braver, T.S., J.R. Gray, G.C. Burgess, and J.N. Towse, *Explaining the many varieties of working memory variation: dual mechanisms of cognitive control*, in *Variation in Working Memory*, A.R.A. Conway, C. Jarrold, M.J. Kane, and A. Miyake, Editors. 2008, Oxford Univ. Press: Oxford, UK. p. 76-106.
- 190. Duncan, J., *An adaptive coding model of neural function in prefrontal cortex*. Nat Rev Neurosci, 2001. **2**(11): p. 820-9.
- 191. Fuster, J.M., *The Prefrontal Cortex*2008, Oxford, UK: Elsevier.
- 192. Crespo-Garcia, M., D. Pinal, J.L. Cantero, F. Diaz, M. Zurron, and M. Atienza, *Working memory processes are mediated by local and long-range synchronization of alpha oscillations*. J Cogn Neurosci, 2013. **25**(8): p. 1343-57.
- 193. Sauseng, P., W. Klimesch, M. Schabus, and M. Doppelmayr, *Fronto-parietal EEG coherence in theta and upper alpha reflect central executive functions of working memory*. Int J Psychophysiol, 2005. **57**(2): p. 97-103.
- 194. Friston, K.J., L. Harrison, and W. Penny, *Dynamic causal modelling*. Neuroimage, 2003. **19**(4): p. 1273-302.
- 195. Stephan, K.E., L.M. Harrison, S.J. Kiebel, O. David, W.D. Penny, and K.J. Friston, *Dynamic causal models of neural system dynamics:current state and future extensions*. J Biosci, 2007. **32**(1): p. 129-44.
- 196. Frazier, T.W., H.A. Demaree, and E.A. Youngstrom, *Meta-analysis of intellectual and neuropsychological test performance in attention-deficit/hyperactivity disorder*. Neuropsychology, 2004. **18**(3): p. 543-55.
- 197. Hart, H., J. Radua, D. Mataix-Cols, and K. Rubia, *Meta-analysis of fMRI studies of timing in attention-deficit hyperactivity disorder (ADHD)*. Neurosci Biobehav Rev, 2012. **36**(10): p. 2248-56.
- 198. Schoechlin, C. and R.R. Engel, *Neuropsychological performance in adult attention-deficit hyperactivity disorder: meta-analysis of empirical data*. Arch Clin Neuropsychol, 2005. **20**(6): p. 727-44.
- 199. Cortese, S., C. Kelly, C. Chabernaud, E. Proal, A. Di Martino, M.P. Milham, and F.X. Castellanos, Toward systems neuroscience of ADHD: a meta-analysis of 55 fMRI studies. Am J Psychiatry, 2012. 169(10): p. 1038-55. PMCID: 3879048
- 200. Norman, L.J., C. Carlisi, S. Lukito, H. Hart, D. Mataix-Cols, J. Radua, and K. Rubia, *Structural and Functional Brain Abnormalities in Attention-Deficit/Hyperactivity Disorder and Obsessive-Compulsive Disorder: A Comparative Meta-analysis*. JAMA Psychiatry, 2016. **73**(8): p. 815-825.
- 201. Bayerl, M., T.F. Dielentheis, G. Vucurevic, T. Gesierich, F. Vogel, C. Fehr, P. Stoeter, M. Huss, and A. Konrad, *Disturbed brain activation during a working memory task in drug-naive adult patients with ADHD*. Neuroreport, 2010. **21**(6): p. 442-6.
- 202. Cubillo, A., A.B. Smith, N. Barrett, V. Giampietro, M. Brammer, A. Simmons, and K. Rubia, *Drug-specific laterality effects on frontal lobe activation of atomoxetine and methylphenidate in attention deficit hyperactivity disorder boys during working memory*. Psychol Med, 2014. **44**(3): p. 633-46.
- 203. Fassbender, C., J.B. Schweitzer, C.R. Cortes, M.A. Tagamets, T.A. Windsor, G.M. Reeves, and R. Gullapalli, *Working memory in attention deficit/hyperactivity disorder is characterized by a lack of specialization of brain function*. PLoS One, 2011. **6**(11): p. e27240. **PMCID**: 3213127
- 204. Hale, T.S., S. Bookheimer, J.J. McGough, J.M. Phillips, and J.T. McCracken, *Atypical brain activation during simple & complex levels of processing in adult ADHD: an fMRI study*. J Atten Disord, 2007. **11**(2): p. 125-40.
- 205. Kobel, M., N. Bechtel, P. Weber, K. Specht, M. Klarhofer, K. Scheffler, K. Opwis, and I.K. Penner, *Effects of methylphenidate on working memory functioning in children with attention deficit/hyperactivity disorder*. Eur J Paediatr Neurol, 2009. **13**(6): p. 516-23.
- 206. Malisza, K.L., J.L. Buss, R.B. Bolster, P.D. de Gervai, L. Woods-Frohlich, R. Summers, C.A. Clancy, A.E. Chudley, and S. Longstaffe, *Comparison of spatial working memory in children with prenatal alcohol exposure and those diagnosed with ADHD; A functional magnetic resonance imaging study*. J Neurodev Disord, 2012. **4**(1): p. 12. **PMCID**: 3436669

- 207. Passarotti, A.M., J.A. Sweeney, and M.N. Pavuluri, *Emotion processing influences working memory circuits in pediatric bipolar disorder and attention-deficit/hyperactivity disorder*. J Am Acad Child Adolesc Psychiatry, 2010. **49**(10): p. 1064-80. **PMCID**: 2957818
- Valera, E.M., S.V. Faraone, J. Biederman, R.A. Poldrack, and L.J. Seidman, *Functional neuroanatomy of working memory in adults with attention-deficit/hyperactivity disorder*. Biol Psychiatry, 2005. **57**(5): p. 439-47.
- 209. Biehl, S.C., K.M. Gschwendtner, A. Guhn, L.D. Muller, S. Reichert, J. Heupel, A. Reif, J. Deckert, M.J. Herrmann, and C.P. Jacob, *Does adult ADHD interact with COMT val (158) met genotype to influence working memory performance?* Atten Defic Hyperact Disord, 2015. 7(1): p. 19-25.
- 210. Mattfeld, A.T., S. Whitfield-Gabrieli, J. Biederman, T. Spencer, A. Brown, R. Fried, and J.D. Gabrieli, Dissociation of working memory impairments and attention-deficit/hyperactivity disorder in the brain. Neuroimage Clin, 2016. **10**: p. 274-82. **PMCID**: PMC4723732
- 211. McCarthy, H., N. Skokauskas, and T. Frodl, *Identifying a consistent pattern of neural function in attention deficit hyperactivity disorder: a meta-analysis*. Psychol Med, 2014. **44**(4): p. 869-80.
- 212. Jaeggi, S.M., M. Buschkuehl, W.J. Perrig, and B. Meier, *The concurrent validity of the N-back task as a working memory measure*. Memory, 2010. **18**(4): p. 394-412.
- 213. Sporns, O., D.R. Chialvo, M. Kaiser, and C.C. Hilgetag, *Organization, development and function of complex brain networks*. Trends Cogn Sci, 2004. **8**(9): p. 418-25.
- 214. Sporns, O., G. Tononi, and G.M. Edelman, *Connectivity and complexity: the relationship between neuroanatomy and brain dynamics*. Neural Netw, 2000. **13**(8-9): p. 909-22.
- 215. Rubinov, M. and O. Sporns, *Complex network measures of brain connectivity: uses and interpretations.* Neuroimage, 2010. **52**(3): p. 1059-69.
- 216. Sporns, O. and R.F. Betzel, *Modular Brain Networks*. Annu Rev Psychol, 2016. **67**: p. 613-40. **PMCID**: PMC4782188
- 217. Peterson, B.S., M.N. Potenza, Z. Wang, H. Zhu, A. Martin, R. Marsh, K.J. Plessen, and S. Yu, *An FMRI study of the effects of psychostimulants on default-mode processing during Stroop task performance in youths with ADHD*. Am J Psychiatry, 2009. **166**(11): p. 1286-94. **PMCID**: PMC3289412
- 218. Karalunas, S.L., H.C. Gustafsson, N.F. Dieckmann, J. Tipsord, S.H. Mitchell, and J.T. Nigg, Heterogeneity in development of aspects of working memory predicts longitudinal attention deficit hyperactivity disorder symptom change. J Abnorm Psychol, 2017. **126**(6): p. 774-792. **PMCID**: PMC5657320
- 219. Keshavan, M.S., S. Vinogradov, J. Rumsey, J. Sherrill, and A. Wagner, *Cognitive training in mental disorders: update and future directions*. Am J Psychiatry, 2014. **171**(5): p. 510-22. **PMCID**: PMC4114156
- 220. Morris, S.E. and B.N. Cuthbert, *Research Domain Criteria: cognitive systems, neural circuits, and dimensions of behavior*. Dialogues Clin Neurosci, 2012. **14**(1): p. 29-37. **PMCID**: PMC3341647
- 221. Insel, T., B. Cuthbert, M. Garvey, R. Heinssen, D.S. Pine, K. Quinn, C. Sanislow, and P. Wang, *Research domain criteria (RDoC): toward a new classification framework for research on mental disorders*. Am J Psychiatry, 2010. **167**(7): p. 748-51.
- 222. Cuthbert, B.N. and M.J. Kozak, *Constructing constructs for psychopathology: the NIMH research domain criteria*. J Abnorm Psychol, 2013. **122**(3): p. 928-37.
- 223. Cuthbert, B.N., *Research domain criteria: toward future psychiatric nosology*. Asian J Psychiatr, 2014. **7**(1): p. 4-5.
- 224. Cuthbert, B.N., *Translating intermediate phenotypes to psychopathology: the NIMH Research Domain Criteria*. Psychophysiology, 2014. **51**(12): p. 1205-6.
- 225. Nigg, J.T., Neuropsychologic theory and findings in attention-deficit/hyperactivity disorder: the state of the field and salient challenges for the coming decade. Biol Psychiatry, 2005. **57**(11): p. 1424-35.
- 226. Mostert, J.C., M. Hoogman, A.M. Onnink, D. van Rooij, D. von Rhein, K.J. van Hulzen, J. Dammers, C.C. Kan, J.K. Buitelaar, D.G. Norris, and B. Franke, *Similar Subgroups Based on Cognitive Performance Parse Heterogeneity in Adults With ADHD and Healthy Controls.* J Atten Disord, 2015. **PMCID**: PMC4884161
- 227. Thaler, N.S., D.T. Bello, and L.M. Etcoff, *WISC-IV profiles are associated with differences in symptomatology and outcome in children with ADHD*. J Atten Disord, 2013. **17**(4): p. 291-301.
- 228. Gomez, R., R.M. Gomez, J. Winther, and A. Vance, *Latent profile analysis of working memory performance in a sample of children with ADHD*. J Abnorm Child Psychol, 2014. **42**(8): p. 1367-79.

- 229. Castellanos, F.X. and E. Proal, *Large-scale brain systems in ADHD: beyond the prefrontal-striatal model.* Trends Cogn Sci, 2012. **16**(1): p. 17-26. **PMCID**: 3272832
- 230. Liston, C., M. Malter Cohen, T. Teslovich, D. Levenson, and B.J. Casey, *Atypical prefrontal connectivity in attention-deficit/hyperactivity disorder: pathway to disease or pathological end point?* Biol Psychiatry, 2011. **69**(12): p. 1168-77.
- 231. Konrad, K. and S.B. Eickhoff, *Is the ADHD brain wired differently? A review on structural and functional connectivity in attention deficit hyperactivity disorder*. Hum Brain Mapp, 2010. **31**(6): p. 904-16.
- 232. Cao, M., N. Shu, Q. Cao, Y. Wang, and Y. He, *Imaging functional and structural brain connectomics in attention-deficit/hyperactivity disorder*. Mol Neurobiol, 2014. **50**(3): p. 1111-23.
- 233. Castellanos, F.X. and Y. Aoki, *Intrinsic Functional Connectivity in Attention-Deficit/Hyperactivity Disorder: A Science in Development*. Biol Psychiatry Cogn Neurosci Neuroimaging, 2016. **1**(3): p. 253-261. **PMCID**: PMC5047296
- 234. De La Fuente, A., S. Xia, C. Branch, and X. Li, *A review of attention-deficit/hyperactivity disorder* from the perspective of brain networks. Front Hum Neurosci, 2013. 7: p. 192. **PMCID**: PMC3654209
- 235. Kasparek, T., P. Theiner, and A. Filova, *Neurobiology of ADHD From Childhood to Adulthood: Findings of Imaging Methods.* J Atten Disord, 2015. **19**(11): p. 931-43.
- 236. Posner, J., C. Park, and Z. Wang, *Connecting the dots: a review of resting connectivity MRI studies in attention-deficit/hyperactivity disorder*. Neuropsychol Rev, 2014. **24**(1): p. 3-15. **PMCID**: PMC4119002
- 237. Rubia, K., A.A. Alegria, and H. Brinson, *Brain abnormalities in attention-deficit hyperactivity disorder: a review*. Rev Neurol, 2014. **58 Suppl 1**: p. S3-16.
- 238. Balanza-Martinez, V., C. Rubio, G. Selva-Vera, A. Martinez-Aran, J. Sanchez-Moreno, J. Salazar-Fraile, E. Vieta, and R. Tabares-Seisdedos, *Neurocognitive endophenotypes (endophenocognitypes) from studies of relatives of bipolar disorder subjects: a systematic review.* Neurosci Biobehav Rev, 2008. 32(8): p. 1426-38.
- 239. Karlsgodt, K.H., P. Bachman, A.M. Winkler, C.E. Bearden, and D.C. Glahn, *Genetic influence on the working memory circuitry: behavior, structure, function and extensions to illness.* Behav Brain Res, 2011. **225**(2): p. 610-22. **PMCID**: PMC3545474
- 240. Lett, T.A., A.N. Voineskos, J.L. Kennedy, B. Levine, and Z.J. Daskalakis, *Treating working memory deficits in schizophrenia: a review of the neurobiology*. Biol Psychiatry, 2014. **75**(5): p. 361-70.
- 241. Wood, R.L. and N.A. Rutterford, *Demographic and cognitive predictors of long-term psychosocial outcome following traumatic brain injury*. J Int Neuropsychol Soc, 2006. **12**(3): p. 350-8.
- Vogt, A., L. Kappos, P. Calabrese, M. Stocklin, L. Gschwind, K. Opwis, and I.K. Penner, *Working memory training in patients with multiple sclerosis comparison of two different training schedules*. Restor Neurol Neurosci, 2009. **27**(3): p. 225-35.
- 243. Westerberg, H., H. Jacobaeus, T. Hirvikoski, P. Clevberger, M.L. Ostensson, A. Bartfai, and T. Klingberg, *Computerized working memory training after stroke--a pilot study*. Brain Inj, 2007. **21**(1): p. 21-9.
- 244. Jones, M.R., B. Katz, M. Buschkuehl, S.M. Jaeggi, and P. Shah, *Exploring N-Back Cognitive Training for Children With ADHD*. J Atten Disord, 2018: p. 1087054718779230. **PMCID**: PMC6445784
- 245. Kofler, M.J., D.E. Sarver, K.E. Austin, H.S. Schaefer, E. Holland, P.A. Aduen, E.L. Wells, E.F. Soto, L.N. Irwin, C. Schatschneider, and C.J. Lonigan, *Can working memory training work for ADHD? Development of central executive training and comparison with behavioral parent training*. J Consult Clin Psychol, 2018. **86**(12): p. 964-979. **PMCID**: PMC6287280
- 246. Schneiders, J.A., B. Opitz, C.M. Krick, and A. Mecklinger, *Separating intra-modal and across-modal training effects in visual working memory: an fMRI investigation*. Cereb Cortex, 2011. **21**(11): p. 2555-64.
- 247. Dahlin, K.I.E., *Working memory training and the effect on mathematical achievement in chidilren with attention deficits and special needs.* Journal of Education and Learning, 2013. **2**(1): p. 118-133.
- 248. Dahlin, E., L. Nyberg, L. Backman, and A.S. Neely, *Plasticity of executive functioning in young and older adults: immediate training gains, transfer, and long-term maintenance.* Psychol Aging, 2008. **23**(4): p. 720-30.
- 249. Backman, L. and L. Nyberg, *Dopamine and training-related working-memory improvement*. Neurosci Biobehav Rev, 2013. **37**(9 Pt B): p. 2209-19.

- 250. Stevens, M.C., *The contributions of resting state and task-based functional connectivity studies to our understanding of adolescent brain network maturation*. Neurosci Biobehav Rev, 2016. **70**: p. 13-32.
- 251. Association, A.P., *Diagnostic and statistical manual of mental disorders*. 4th ed1994, Washington, DC: American Psychiatric Association.
- 252. Kaufman, J., B. Birmaher, D. Brent, U. Rao, C. Flynn, P. Moreci, D. Williamson, and N. Ryan, *Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data.* J Am Acad Child Adolesc Psychiatry, 1997. **36**(7): p. 980-8.
- 253. Achenbach, T.M. and C. Edelbrock, *Manual of the Child Behavior Checklist and Revised Child Behavior Profile*1983, Burlington: University of Vermont, Department of Psychiatry.
- 254. Conners, C.K., Conners 3, 2008, Multi-Health Systems, Inc.
- 255. Weiss, M., The unique apsective of assessment in ADHD. Primary Psychiatry, 2010. 17(5): p. 21-25.
- 256. Gullone, E. and K. Robinson, *The inventory of parent and peer attachment revised (IPPA-R) for Children: A psychometric investigation*. Clinical Psychology and Psychotherapy, 2005. **12**: p. 67-79.
- 257. Beck, A.T., R.A. Steer, and G.K. Brown, *Beck Depression Inventory—II (BDI–II)*1996, San Antonio, TX: Harcourt Assessment, Inc.
- 258. March, J.S., Multidimensional Anxiety Scale for Children (2nd Edition).
- 259. Moberg, D.P., Screening for Alcohol and Other Drug Problems using the Adolescent Alcohol and Drug Involvement Scale (AADIS), 2005, University of Wisconsin Medical School: Center for Health Policy and Program Evaluation.
- 260. Fagerstrom, K.O. and N.G. Schneider, *Measuring nicotine dependence: a review of the Fagerstrom Tolerance Questionnaire*. J Behav Med, 1989. **12**(2): p. 159-82.
- 261. Petersen, A.C., L. Crockett, and M. Richards, *A self-report measure of pubertal status: Reliability, Validity, and Initial Norms.* Journal of Youth and Adolescence, 1988. **17**: p. 117-133.
- 262. Annett, M., *A classification of hand preference by association analysis*. British Journal of Psychology, 1970. **61**: p. 303-321.
- 263. Hollingshead, A., *The four-factor index of social status*1975, New Haven, CT: Unpublised manuscript, Yale University.
- 264. Sitskoorn, M.M., A. Aleman, S.J. Ebisch, M.C. Appels, and R.S. Kahn, *Cognitive deficits in relatives of patients with schizophrenia: a meta-analysis*. Schizophrenia Research, 2004. **71**(2-3): p. 285-95.
- 265. Corporation, P., Wechsler Intelligence Scale for Children (4th Edition)1999, San Antonio, TX: Harcourt Assessment, Inc.
- 266. Leung, H.C., H. Oh, J. Ferri, and Y. Yi, *Load response functions in the human spatial working memory circuit during location memory updating*. Neuroimage, 2007. **35**(1): p. 368-77.
- 267. Conners, C.K., *Conners' Continuous Performance Test II*2005: Psychological Assessment Resources, Inc.
- 268. <a href="http://www.cogstate.com/">http://www.cogstate.com/</a>.
- 269. Lewis, P.A. and R.C. Miall, *Brain activation patterns during measurement of sub- and supra-second intervals*. Neuropsychologia, 2003. **41**(12): p. 1583-92.
- 270. Wöstmann, N.M., D.S. Aichert, A. Costa, K. Rubia, H.-J. Möller, and U. Ettinger, *Reliability and plasticity of response inhibition and interference control*. Brain and Cognition, 2013. **81**(1): p. 82-94.
- 271. Wechsler, D., *Wechsler Abbreviated Scale of Intelligence*, 1999, The Psychological Corporation: Harcourt Brace & Company: New York, NY.
- 272. Eich, T.S., D.E. Nee, C. Insel, C. Malapani, and E.E. Smith, *Neural Correlates of Impaired Cognitive Control over Working Memory in Schizophrenia*. Biol Psychiatry, 2013.
- 273. Murty, V.P., F. Sambataro, E. Radulescu, M. Altamura, J. Iudicello, B. Zoltick, D.R. Weinberger, T.E. Goldberg, and V.S. Mattay, *Selective updating of working memory content modulates meso-cortico-striatal activity*. Neuroimage, 2011. **57**(3): p. 1264-72. **PMCID**: PMC3908780
- 274. Van Essen, D.C., K. Ugurbil, E. Auerbach, D. Barch, T.E. Behrens, R. Bucholz, A. Chang, L. Chen, M. Corbetta, S.W. Curtiss, S. Della Penna, D. Feinberg, M.F. Glasser, N. Harel, A.C. Heath, L. Larson-Prior, D. Marcus, G. Michalareas, S. Moeller, R. Oostenveld, S.E. Petersen, F. Prior, B.L. Schlaggar, S.M. Smith, A.Z. Snyder, J. Xu, E. Yacoub, and W.U.-M.H. Consortium, *The Human Connectome Project: a data acquisition perspective*. Neuroimage, 2012. 62(4): p. 2222-31. PMCID: 3606888

- 275. Marcus, D.S., J. Harwell, T. Olsen, M. Hodge, M.F. Glasser, F. Prior, M. Jenkinson, T. Laumann, S.W. Curtiss, and D.C. Van Essen, *Informatics and data mining tools and strategies for the human connectome project*. Front Neuroinform, 2011. **5**: p. 4. **PMCID**: 3127103
- 276. Jenkinson, M., C.F. Beckmann, T.E. Behrens, M.W. Woolrich, and S.M. Smith, *Fsl.* Neuroimage, 2012. **62**(2): p. 782-90.
- 277. Rao, U., C. Hammen, and S.E. Daley, *Continuity of depression during the transition to adulthood: a 5-year longitudinal study of young women.* J Am Acad Child Adolesc Psychiatry, 1999. **38**(7): p. 908-15.
- 278. Glasser, M.F., T.S. Coalson, E.C. Robinson, C.D. Hacker, J. Harwell, E. Yacoub, K. Ugurbil, J. Andersson, C.F. Beckmann, M. Jenkinson, S.M. Smith, and D.C. Van Essen, *A multi-modal parcellation of human cerebral cortex*. Nature, 2016. **536**(7615): p. 171-8. **PMCID**: PMC4990127
- 279. Ji, J.L., M. Spronk, K. Kulkarni, G. Repovs, A. Anticevic, and M.W. Cole, *Mapping the human brain's cortical-subcortical functional network organization*. Neuroimage, 2019. **185**: p. 35-57. **PMCID**: PMC6289683
- 280. Dosenbach, N.U.F., J.M. Koller, E.A. Earl, O. Miranda-Dominguez, R.L. Klein, A.N. Van, A.Z. Snyder, B.J. Nagel, J.T. Nigg, A.L. Nguyen, V. Wesevich, D.J. Greene, and D.A. Fair, *Real-time motion analytics during brain MRI improve data quality and reduce costs*. Neuroimage, 2017. **161**: p. 80-93. **PMCID**: 5731481
- 281. Griffanti, L., G. Salimi-Khorshidi, C.F. Beckmann, E.J. Auerbach, G. Douaud, C.E. Sexton, E. Zsoldos, K.P. Ebmeier, N. Filippini, C.E. Mackay, S. Moeller, J. Xu, E. Yacoub, G. Baselli, K. Ugurbil, K.L. Miller, and S.M. Smith, *ICA-based artefact removal and accelerated fMRI acquisition for improved resting state network imaging*. Neuroimage, 2014. **95**: p. 232-47. **PMCID**: PMC4154346
- 282. Salimi-Khorshidi, G., G. Douaud, C.F. Beckmann, M.F. Glasser, L. Griffanti, and S.M. Smith, *Automatic denoising of functional MRI data: combining independent component analysis and hierarchical fusion of classifiers.* Neuroimage, 2014. **90**: p. 449-68. **PMCID**: PMC4019210
- 283. Bullmore, E. and O. Sporns, *Complex brain networks: graph theoretical analysis of structural and functional systems.* Nat Rev Neurosci, 2009. **10**(3): p. 186-98.
- 284. Telesford, Q.K., S.L. Simpson, J.H. Burdette, S. Hayasaka, and P.J. Laurienti, *The brain as a complex system: using network science as a tool for understanding the brain.* Brain Connect, 2011. **1**(4): p. 295-308. **PMCID**: PMC3621511
- 285. Power, J.D., B.L. Schlaggar, and S.E. Petersen, *Recent progress and outstanding issues in motion correction in resting state fMRI*. Neuroimage, 2015. **105**: p. 536-51. **PMCID**: PMC4262543
- 286. Power, J.D., K.A. Barnes, A.Z. Snyder, B.L. Schlaggar, and S.E. Petersen, *Steps toward optimizing motion artifact removal in functional connectivity MRI; a reply to Carp.* Neuroimage, 2013. **76**: p. 439-41. **PMCID**: 3834590
- 287. Smith, S.M., D. Vidaurre, C.F. Beckmann, M.F. Glasser, M. Jenkinson, K.L. Miller, T.E. Nichols, E.C. Robinson, G. Salimi-Khorshidi, M.W. Woolrich, D.M. Barch, K. Uğurbil, and D.C. Van Essen, *Functional connectomics from resting-state fMRI*. Trends in Cognitive Sciences, 2013. **17**(12): p. 666-682.
- 288. Brehmer, Y., A. Rieckmann, M. Bellander, H. Westerberg, H. Fischer, and L. Backman, *Neural correlates of training-related working-memory gains in old age*. Neuroimage, 2011. **58**(4): p. 1110-20.
- 289. Fisher, M., C. Holland, M.M. Merzenich, and S. Vinogradov, *Using neuroplasticity-based auditory training to improve verbal memory in schizophrenia*. Am J Psychiatry, 2009. **166**(7): p. 805-11. **PMCID**: PMC2720319
- 290. Fisher, M., C. Holland, K. Subramaniam, and S. Vinogradov, *Neuroplasticity-based cognitive training in schizophrenia: an interim report on the effects 6 months later*. Schizophr Bull, 2010. **36**(4): p. 869-79. **PMCID**: PMC2894606
- 291. Charvet, L.E., M. Kasschau, A. Datta, H. Knotkova, M.C. Stevens, A. Alonzo, C. Loo, K.R. Krull, and M. Bikson, *Remotely-supervised transcranial direct current stimulation (tDCS) for clinical trials:* guidelines for technology and protocols. Front Syst Neurosci, 2015. **9**: p. 26. **PMCID**: PMC4362220
- 292. Knotkova H, C.A., Stevens M, Riggs A, Charvet L, Bikson M. . In: (eds): . , in progress., *Home-based patient-delivered remotely supervised tDCS. Chapter 14*, in *Practical Guide to Transcranial Direct Current Stimulation*, H. Knotkova, M.A. Nitsche, M. Bikson, and A.J. Woods, Editors. in progress, Springer Publishing.
- 293. Little, R. and D. Rubin, Statistical analysis with missing data2002, New York: Wiley.

- 294. Allison, P. *Handling missing data by maximum likelihood*. Statistics and Data Analysis: SAS Global Forum, 2012.
- 295. Enders, C.K., *Applied missing data analysis* 2010, New York: Guilford Press.
- 296. Wilcox, R.R., *Introduction to robust estimation and hypothesis testing* 2012, New York: Academic Press.
- 297. Winkler, A.M., G.R. Ridgway, M.A. Webster, S.M. Smith, and T.E. Nichols, *Permutation inference for the general linear model*. Neuroimage, 2014. **92**: p. 381-97. **PMCID**: 4010955
- 298. Lachin, J.M., J.P. Matts, and L.J. Wei, *Randomization in clinical trials: conclusions and recommendations*. Control Clin Trials, 1988. **9**(4): p. 365-74.
- 299. Wei, L.J. and J.M. Lachin, *Properties of the urn randomization in clinical trials*. Control Clin Trials, 1988. **9**(4): p. 345-64.
- 300. Jo, B., E.M. Ginexi, and N.S. Ialongo, *Handling missing data in randomized experiments with noncompliance*. Prev Sci, 2010. **11**(4): p. 384-96. **PMCID**: 2912956
- 301. Dovis, S., M. Maric, P.J.M. Prins, and S. Van der Oord, *Does executive function capacity moderate the outcome of executive function training in children with ADHD?* Atten Defic Hyperact Disord, 2019. **11**(4): p. 445-460.
- 302. Matysiak, O., A. Kroemeke, and A. Brzezicka, *Working Memory Capacity as a Predictor of Cognitive Training Efficacy in the Elderly Population*. Front Aging Neurosci, 2019. **11**: p. 126. **PMCID**: PMC6554703
- 303. van der Donk, M.L., A.C. Hiemstra-Beernink, A.C. Tjeenk-Kalff, A. van der Leij, and R.J. Lindauer, Predictors and Moderators of Treatment Outcome in Cognitive Training for Children With ADHD. J Atten Disord, 2016.
- 304. Durston, S., J. van Belle, and P. de Zeeuw, *Differentiating frontostriatal and fronto-cerebellar circuits in attention-deficit/hyperactivity disorder*. Biol Psychiatry, 2011. **69**(12): p. 1178-84.
- 305. Nigg, J.T. and B.J. Casey, *An integrative theory of attention-deficit/ hyperactivity disorder based on the cognitive and affective neurosciences*. Dev Psychopathol, 2005. **17**(3): p. 785-806.
- 306. Sagvolden, T., E.B. Johansen, H. Aase, and V.A. Russell, *A dynamic developmental theory of attention-deficit/hyperactivity disorder (ADHD) predominantly hyperactive/impulsive and combined subtypes*. Behav Brain Sci, 2005. **28**(3): p. 397-419; discussion 419-68.